# Traumed - C1502

Multi-centre, Double-blind, Randomised, Active- and Placebo-Controlled, Confirmatory Trial to Demonstrate Efficacy and Safety of Traumed® Gel in Patients having Acute Ankle Sprain

# STATISTICAL ANALYSIS PLAN (SAP)

Study code C1502

Study Protocol 03.02.2020, Final Version 4.0

Study design Randomised, double-blind, active- and placebo-controlled

confirmatory clinical trial

Sponsor /contract party Biologische Heilmittel Heel GmbH

Dr.-Reckeweg-Straße 2-4 D-76532 Baden-Baden

Germany

# SAP Revision History

| Version | Date | Author | Review | Comments |
|---|---|---|---|---|
| Draft 1.0 | 07.12.2018 | J.C. Vester | V.W. Rahlfs | Initial Draft |
| Draft-to-<br>Final 1.0 | 12.04.2021 | J.C. Vester | V.W. Rahlfs | Adaption to Amendment to Protocol version 3.0 (Protocol version 4.0) Implementation of final BDRM Decisions |
| Final 1.0 | 20.04.2021 | J.C. Vester | V.W. Rahlfs | Switch to American English (AE) Additional operationalization in section 9.4.2. Stratification Individual Dataset Assignment in Section 13.2 |

### CONFIDENTIAL

THIS SAP CONTAINS CONFIDENTIAL INFORMATION OF IDV AND BIOLOGISCHE HEILMITTEL HEEL GMBH AND IS INTENDED SOLELY FOR THE PURPOSE OF THIS STUDY. THIS SAP MAY NOT BE DISCLOSED TO PARTIES NOT ASSOCIATED WITH THIS STUDY FOR ANY PURPOSE WITHOUT WRITTEN CONSENT OF IDV AND BIOLOGISCHE HEILMITTEL HEEL GMBH.

# 1. SIGNATURES

Trial Statistician(s)

20.04.2021

date

Prof. Johannes C. Vester

IDV Data Analysis and Study Planning, Gauting, Germany

Review:

20.4.2021

date

Dr. Volker W. Rahlfs CStat (RSS)

IDV Data Analysis and Study Planning, Gauting, Germany

# SAP Approval Sponsor's Representative

21 April 2021

date

Dr Christine Frank, PhD

Senior Clinical Project Manager Biologische Heilmittel Heel GmbH, Baden-Baden, Germany

# SAP Approval National Coordinating Investigator

22.04.21

date



Prof. Dr. med. Thomas Becker, MD

Universitätsklinikum Schleswig-Holstein Director Klinik für Allgemeine, Viszeral-, Thorax-, Transplantations- und Kinderchirurgie Kiel, Germany SAP Approval Scie

22421

date



Prof. Dr. med. Ludger Gerdesmeyer, MD, PhD

Universitätsklinikum Schleswig-Holstein Chairman Sektion für Onkologische und Rheumatologische Orthopädie Kiel, Germany

# 2. TABLE OF CONTENTS

| 1. | Signatures | 2 |
|---|---|---|
| 2. | Table of Contents | 6 |
| 3. | Preliminary Remarks | 8 |
| 4. | Abbreviations | 9 |
| 5. | Introduction | 11 |
| 5/5 | 5.1 Background information | |
| 6. | Excerpts from Final Protocol | |
| • | 6.1 Protocol Synopsis | |
| | 6.2 Schedule of Study Procedures | |
| | 6.3 Assessment of Efficacy | |
| | 6.3.1 Primary Efficacy Parameter | |
| | 6.3.2 Secondary Efficacy Parameters | |
| | 6.3.3 Safety Assessments | 23 |
| 7. | Blind Data Transfers and Quality Assurance | 24 |
| 8. | Changes to the Protocol | |
| 9. | Additional Specifications to the Protocol | |
| | 9.1 Standard Procedures | |
| | 9.2 Demography and Baseline Characteristics | |
| | 9.2.1 Operationalizations in Final Protocol | |
| | 9.2.2 Additional Operationalizations | |
| | 9.3 Evaluations and Endpoints – First Line Analysis | |
| | 9.3.1 Primary Efficacy Variable | |
| | 9.3.1.1 Operationalizations in Final Protocol | |
| | 9.3.1.2 Additional Operationalizations | 29 |
| | 9.3.2 Secondary Efficacy Variables | |
| | 9.3.2.1 Operationalizations in Final Protocol | |
| | 9.3.2.2 Additional Operationalizations | |
| | 9.4 Evaluations and Endpoints – Second Line Analysis | |
| | 9.4.1 Nonparametric Analysis | |
| | 9.4.1.1 Operationalizations in Final Protocol | |
| | 9.4.1.2 Additional Operationalizations | |
| | 9.4.2 Stratification | |
| | 9.4.2.1 Operationalizations in Final Protocol 9.4.2.2 Additional Operationalizations | |
| | 9.5 Accounting for Missing Data | |
| | 9.5.1.1 Operationalizations in Final Protocol | |
| | 9.5.1.2 Additional Operationalizations | |
| | 9.6 Evaluations and Endpoints – Safety | |
| | 9.6.1.1 Operationalizations in Final Protocol | |
| | 9.6.1.2 Additional Operationalizations | |
| | 9.7 Analysis Populations | 36 |
| | 9.7.1.1 Operationalizations in Final Protocol | |
| | 9.7.1.2 Additional Operationalizations | 37 |

| 10. | Softwar | e Applied | 38 |
|-----|----------|---------------------------------------------------|----|
| 11. | Post ho | c Changes to Planned Analyses (Post Unblinding) | 38 |
| 12. | Referen | ices | 39 |
| 13. | Append | lix | 44 |
| | 13.1 BE | DRM Decisions | 44 |
| | 13.1.1 | Problem Cases | 44 |
| | | Other Decisions | |
| | 13.2 Inc | dividual Dataset Assignment | 44 |
| | | ble of Contents for Data Displays (Items of eCRF) | |
| | 13.3.1 | Tables | |
| | 13.3.2 | Listings | 69 |
| | 13.3.3 | Figures | 71 |
| | 13.4 Cli | inical Trial Report (CTR) Specifications | 73 |
| | 13.4.1 | Core CTR Specifications | 73 |
| | 13.4.2 | Appendices: | 73 |

### 3. PRELIMINARY REMARKS

The C1502 Statistical Analysis Plan (SAP) is a detailed technical extension to the C1502 Study Protocol Version 3.0 (1 December 2017), following principles of the Guidelines ICH E3/E6R2/E9, as well as relevant IDV SOPs and/or guidelines as far as applicable to the trial. This plan describes the statistical analysis planned to be performed after all enrolled patients data are available for evaluation. This Statistical Analysis Plan will be finalized and signed after raw database hard lock, but before generation of the final analysis database as well as before unblinding approval. Formal records will be kept of when the Statistical Analysis Plan was finalized as well as when the blind was subsequently broken.

All planned analyses identified in this SAP will be included in the Clinical Trial Report (CTR). Exploratory analyses not necessarily identified in this SAP may be performed to support planned analyses. Any *post-hoc* or unplanned analyses not specified in this SAP will be clearly identified as such in the CTR.

The following documents were reviewed when preparing this SAP:

- C1502 Study Protocol Version 4.0 (3 February 2020)
- Amendment Summary Document for Substantial protocol Changes (3 February 2020)
- HE13226\_eCRF Specification\_v3.0\_20180425
- 20210113 C1502 Issue Overview FINAL
- C1502 MTG NOTES BDRM 09MAR2021 20210324 (Blind Data Review Meeting)
- C1502\_LIVE17\_Risk Based Centralized Statistical Monitoring\_IDV\_20210409 (Hardlock)

Readers of this SAP are encouraged to read the Clinical Trial protocol for details on the conduct of this clinical trial and the operational aspects of clinical assessments and timing for completing a patient in this trial.

# 4. ABBREVIATIONS

| Abbreviation | Definition |
|---|---|
| ADL | Activities of Daily Living |
| AR(s) | Adverse Reaction(s) |
| AE(s) | Adverse Event(s) |
| ANCOVA | Analysis of covariance |
| AUC | Area under the curve |
| BDRM | Blind Data Review Meeting |
| BMI | Body Mass Index |
| С | Celsius degree |
| CCSI | Company Core Safety Information |
| CI | confidence interval |
| CMH | Cochran-Mantel-Haenszel (pooling) |
| COX-2 | Cyclooxygenase type 2 |
| CRO | Contract Research Organisation |
| CStat | Chartered Statistician |
| eCRF | electronic Case Report Form |
| EMA | European Medicines Agency |
| ЕоТ | End of Treatment |
| EU | European Union |
| FAAM | Foot and Ankle Ability Measure |
| FAS | Full analysis set |
| GCP | Good Clinical Practice |
| GMDS | Deutsche Gesellschaft für Medizinische Informatik, Biometrie und |
| | Epidemiologie e.V. |
| GMP | Good Manufacturing Practice |
| HSPC | high security PC (personal computer) |
| ICH | International Conference on Harmonisation |
| IEC | Independent Ethics Committee |
| IL | Interleukin |
| IMP | Investigational Medicinal Product |
| ITT | Intent-to-treat |
| IUD | Intrauterine device |
| IUS | Intrauterine hormone-releasing system |
| LOCF | Last Observation Carried Forward |
| LPCP | Last Percentile Carried Forward |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | Milligram |
| mg/d | Milligrams per day |
| mm | Millimeter |
| MMRM | mixed-effect models for repeated measures |
| MW | Mann-Whitney |
| N | Number of patients |
| 11 | ivamori of patients |

| Abbreviation | Definition |
|---------------------------|----------------------------------------|
| NI | Non-inferiority |
| NSAID | Non-steroidal anti-inflammatory drug |
| PP | Per protocol |
| PRN | When necessary (pro re nata) |
| QPPV | Qualified person for pharmacovigilance |
| RICE | Rest, Ice, Compression and Elevation |
| RSS | Royal Statistical Society |
| SAE(s) | Serious Adverse Event(s) |
| SAP | Statistical Analysis Plan |
| SD | standard deviation |
| SOC | Summary Of Changes |
| SOP | Standard Operating Procedure |
| SmPC | Summary of Product Characteristics |
| TGF-β | transforming growth factor beta |
| TNF-α | tumor necrosis factor alpha |
| VAS | Visual Analog Scale |
| VASPM | Pain score on passive movement (VAS) |
| WMA | World Medical Assembly |
| WMW Wilcoxon-Mann-Whitney | |

### 5. INTRODUCTION

# 5.1 Background information

Ankle sprain injuries are the most common type of joint sprain. The prevalence of ankle joint sprains accounts for 21% of joint injuries in the body. Although somewhat rare, high-ankle or syndesmotic ankle sprains occur in up to 15% of ankle traumas (Childs, 2012).

Lateral ankle sprains are the most prevalent musculoskeletal injury in physically active populations. They also have a high prevalence in the general population and pose a substantial healthcare burden. The injury mechanism is characterised by a high velocity inversion and internal rotation of the ankle/foot complex. The treatment for acute lateral ankle sprain is quite variable, with many patients returning to activity in a short period of time; however, half of the population may never seek initial care (Gribble et al. 2016). Inadequate treatment of ankle sprains can lead to chronic problems such as decreased range of motion, pain, and joint instability (Wolfe et al. 2001; Ivins et al. 2006).

Many patients who suffer from some form of ankle injury do not seek treatment, as a treatment regimen would significantly impact their physical activities, such as training, practicing and competing for a substantial period of time (McKay et al. 2001). A study (Hubbard et al. 2009) showed that natural recovery from ankle sprain takes longer than 8 weeks – a significant time for any athlete to be away from activity.

Some evidence suggests that previous injuries or limited joint flexibility may contribute to ankle sprains. The initial assessment of an acute ankle injury should include questions about the timing and mechanism of the injury. Ankle sprains can be classified as grade 1, grade 2 or grade 3, depending on the severity of the injury (Wexler et al. 1998).

Physicians should apply e.g. the Ottawa ankle rules to determine whether radiography is needed. According to the Ottawa criteria, radiography is indicated if there is pain in the malleolar or midfoot zone, and either bone tenderness over an area of potential fracture (i.e. lateral malleolus, medial malleolus, base of fifth metatarsal, or navicular bone) or an inability to bear weight for four steps immediately after the injury and in the emergency department or physician's office (Tiemstra, 2012).

Clinically, a first approach to soft tissue injuries follows the RICE principle (simultaneous combination of all 4 elements Rest, Ice, Compression and Elevation). The objective of RICE is to stop the injury-induced bleeding into the muscle tissue and thereby minimize the extent of the injury.

In a study in acute ankle sprain, an accelerated intervention with early therapeutic exercise during the first week after ankle sprain improved ankle function compared with RICE, although the groups did not differ at any other time point for pain at rest, pain on activity, or swelling (Bleakley et al. 2010).

Controlled trials of non-steroidal anti-inflammatory drugs (NSAIDs) e.g. diclofenac, piroxicam, celecoxib, naproxen and others in patients with ankle sprain showed that

compared with placebo, NSAIDs were associated with improved pain control and function, decreased swelling, and more rapid return to activity. To reduce or even avoid the well-known side effects of systemic NSAIDs topical application is an efficacious alternative (Lin et al. 2004, Mason et al. 2001, Mason et al. 2004, Heumann Pharma, Predel et al. 2004).

Reviews of diclofenac have consistently demonstrated its efficacy in reducing pain and inflammation in acute and chronic conditions compared with placebo. Diclofenac is meanwhile considered to be the gold standard in the treatment of joint sprains and other conditions. Topical diclofenac is well tolerated and is associated with fewer side-effects than other topical NSAIDs, mostly mild, easily resolved local skin irritation (Banning 2008, Zacher et al. 2008, Simon et al. 2009). A systematic review and meta-analysis of blinded, randomized, placebo-, vehicle- or active-controlled trials concluded that topical diclofenac appears to be generally well tolerated for cutaneous use in acute and chronic musculoskeletal conditions (Taylor et al. 2011). For these reasons, diclofenac gel was chosen as a comparator for this trial.

Traumeel® is a German non-prescription drug sold for more than 50 years over the counter in pharmacies in Germany, Austria, Switzerland and in more than 50 other countries worldwide in the form of oral drops, tablets, ointment and ampoules. A gel formulation of the product is available in Austria, Belgium, The Netherlands, Poland and Spain in the EU, and in some other countries worldwide for human use as Traumeel® gel. In Germany the gel variant of the product is planned to be submitted for authorization as Traumed® gel.

Traumeel® (for topical application, either as ointment or a gel) is produced in accordance with the German Homeopathic Pharmacopoeia and the European Pharmacopoeia. quality of Traumed<sup>®</sup> gel is guaranteed both by the use of active substances and excipients that meet the requirements of the Homeopathic Pharmacopoeia and the European Pharmacopoeia and by production in accordance with good manufacturing practice (GMP) guidelines. Local tolerability data of Traumeel® gel are available from a local tolerability trial. Traumeel® is a fixed combination of plant and mineral extracts used for treating inflammation and pain caused by musculoskeletal injuries (Schneider, 2011). Efficacy and tolerability of Traumeel® for musculoskeletal injuries have been reported in randomized controlled trials, which demonstrate reductions in pain and swelling, and improvements in the mobility of joints such as ankle and knee (Zell et al. 1998, Böhmer et al. 1992, Thiel et al. 1994). Traumeel® has proven efficacy which is equivalent to conventional management (Schneider et al. 2008), NSAIDs (Birnesser et al. 2004) and to diclofenac (Schneider et al. 2005) in pain relief and improving joint mobility. Traumeel® is well tolerated, with very few adverse effects (Arora et al 2000, Birnesser et al. 2004, Böhmer et al. 1992, Thiel et al. 1994, Schneider et al. 2005. Schneider et al. 2008, Zenner et al. 1992, Zenner et al. 1994, Zenner et al. 1997).

Evidence for the inflammation regulating action of Traumeel® comes from Porozov et al. 2004 who conducted a study to evaluate the effect of Traumeel® on human leukocyte function. Specifically, the action of Traumeel® was studied on activated human T-cells,

monocytes and gut epithelial cells in terms of its effect on the pro-inflammatory mediators IL-1 $\beta$  (interleukin-1 $\beta$ ), TNF- $\alpha$  (tumor necrosis factor- $\alpha$ ) and IL-8 (interleukin-8) *in vitro*.

The researchers found that Traumeel® modulates the secretion of IL-1β, TNF-α and IL-8 in resting as well as in activated immune cells. It was observed that T-cell and monocyte proliferation was not affected. The researchers concluded that Traumeel® reduces pro-inflammatory cytokines in resting and activated immunocytes *in vitro*, as well as in resting and activated colon epithelial cells, suggesting that the first-line and mobile arm of immune defence is activated by Traumeel®. The study concluded that the results support the characterization of Traumeel® as an inflammation-regulating medication.

Traumeel® acts differently to NSAIDs, its anti- inflammatory effect results from the synergistic interaction between its components on the different phases of the inflammatory response (Lussignoli et al. 1999).

In vitro studies (Wexler et al. 1998) showed that the ingredients of Traumeel® are non-cytotoxic to granulocytes, lymphocytes, platelets and endothelial cells, indicating that the normal defensive and homeostatic functions of these cells are preserved during treatment with Traumeel®. Additional data alluding to the mode of action of Traumeel® comes from basic research (Heine et al. 2002) which has shown that the organic components of Traumeel® stimulate lymphocytes to synthesize and secrete the cytokine TGF-β (transforming growth factor-β) in whole blood cultures. TGF-β reduces pro-inflammatory substances such as TNF-α, Interferon-gamma, IL-1 and IL-2.

Traumeel<sup>®</sup> seems to modulate the healing process to assist resolution of symptoms including pain.

For homeopathic substances, pharmacokinetic investigations are not relevant regarding the efficacy of a substance or a combination of different substances. An expert's opinion on toxicology states that the material available and clinical experience provides no indication of toxicological risks associated with ingredients of the homeopathic drug Traumeel® when the product is applied as recommended.

A Traumeel® ointment and gel non-inferiority clinical trial (TAASS; Gonzalez et al. 2013) was conducted in 449 athletes with grade 1 or grade 2 acute ankle sprain as a multi-center, randomized, blinded, parallel-group, active controlled clinical trial.

The baseline medians of the pain Visual Analog Scale (VAS) scale were lying between 52.6 mm and 55.7 mm (minimum 29.9 mm, maximum 94.8 mm). All groups showed strong pain decrease with a final median of 0 mm (total pain relief) after 6 weeks. At the primary endpoint day 7 the median was 21.6 (Traumeel® ointment), 16.0 (Traumeel® Gel) and 17.5 (diclofenac gel).

Total pain relief at day 7 (-100.0%) was reached in 8.5% of the patients in the Traumeel® ointment group, in 5.0% of the patients in the Traumeel® gel group and in 5.9% of the patients in the diclofenac gel group.

The baseline medians of the Foot and Ankle Ability Measure (FAAM) Activities of daily living (ALD) score were lying between 51.2 and 56.0 (minimum 2.4, maximum 98.3). All groups showed strong increase of FAAM-ADL with a final median of 100 (best score) after 6 weeks. At the primary endpoint day 7 the median was 81.0 (Traumeel® ointment), 85.1 (Traumeel® gel) and 79.8 (diclofenac gel). Thus, the best median score was observed in the Traumeel® gel group, followed by the Traumeel® ointment group and the diclofenac gel group.

Altogether, 31 out of 447 patients of the safety population (6.9%) suffered from 43 AEs. At least one AE was experienced by 9 patients out of 152 patients (5.9%) of the Traumeel® ointment group, by 14 patients out of 148 patients (9.5%) of the Traumeel® Gel group and by 8 patients out of 147 patients (5.4%) of the diclofenac gel group. The proportion of treated patients with AEs was therefore below 10% in all treatment groups. The most common AE was headache, reported in 13 cases. None of these 13 headaches was assessed by the investigator as "possible" or "probable" related to investigational medication. Serious AEs were experienced by no patient and in no treatment group. There were no serious or fatal AEs.

Pharmacovigilance data on Traumeel® Gel show 9 non-serious Adverse Reactions (ARs), assessed with "possible" or "probable" causal relationship to the treatment, in the time period between 01.01.2008 and 01.01.2016. Two of the cases reporting skin reactions were received from a clinical trial (TRS-ESP/ TAASS trial/ EudraCT number: 2008-007939-4). One case reported eye hypersensitivity symptoms and can be considered as an isolated case. The other cases related to hypersensitivity skin conditions, which are already listed in the respective label (allergic reactions). The units sold on Traumeel® gel during this period are 2.047.579 packages. Thus, the incidence ratio for the non-serious ADRs is 7 cases per 2.047.579 packages, which means an event rate of 1:292.511.

No AEs indicative of Traumeel® overdose, either for ointment or gel, have been reported. Based on the available data, the overall safety profile of Traumeel® medications is considered being very good.

According to the SmPC of Diclofenac Heumann Gel (HEUMANN PHARMA GMBH & CO. GENERICA KG, N., 2013) its use is contraindicated in case of sensitivity to any components of the gel (e.g. paracetamol, isopropanol, ethanol; see [protocol] section 6.1.1 for description of other ingredients), for patients in whom asthma attacks, skin rash or acute rhinitis are triggered by acetylsalicylic acid or NSAIDs, treatment for open wound, infections or inflammation of the skin (e.g. eczema) or application on the mucosa. Possible side effects are also described in the SmPC.

Diclofenac Heumann Gel is only recommended in first and second trimester of pregnancy if absolutely required. Systemic administration of diclofenac inhibited the ovulation in rabbits and the implantation and embryogenesis in rats. Teratogenicity was investigated in rats, cats and rabbits. Based on the available non-clinical data, diclofenac is considered non-teratogenic. (HEUMANN PHARMA GMBH & CO. GENERICA KG, N., 2013).

Placebo is contraindicated in case of sensitivity to any components of the gel, see [protocol] section 6.1.1 for description.

In the TAASS trial (Gonzalez et al. 2013) topical treatment with Traumeel® or diclofenac resulted in reduction of pain and restoration of function in patients with grade 1 or grade 2 ankle sprain. The current trial is designed to demonstrate the superior efficacy of Traumed® gel versus placebo and to assess the non-inferiority of Traumed® gel compared to diclofenac gel.

### 6. EXCERPTS FROM FINAL PROTOCOL

### 6.1 Protocol Synopsis

| Sponsor:<br>Biologische Heilmittel Heel<br>GmbH | Name of Medical Product:<br>Traumed <sup>®</sup> Gel | Active Ingredient(s): Homeopathic preparation, containing herbal and mineral ingredients as described in the Clinical Study Protocol |
|---|---|---|
| EudraCT number: 2016-00479 | 92-50 | Indication: Acute ankle sprain |

### Study Title:

Multi-centre, Double-blind, Randomised, Active- and Placebo-Controlled, Confirmatory Trial to Demonstrate Efficacy and Safety of Traumed® Gel in Patients having Acute Ankle Sprain

### Study Sites:

Multi-centre study in Germany (at approximately 35 sites, trauma centres (surgeons), emergency units, sport medicine practices (physicians), general practitioners

Coordinating Investigator: Prof Dr med Thomas Becker

Universitätsklinikum Schleswig-Holstein

Arnold Heller Straße 3

24105 Kiel Germany

Phone: +49 431 5002 4485

**Study Duration:** 

February 2018

Ш

Study Phase:

First patient first visit:

Last patient last visit planned:

December 2020

### Study objectives:

The primary objective of the study is to demonstrate the superior efficacy of Traumed® gel versus placebo in patients with acute lateral ankle sprain

The secondary objectives are:

- · to assess non-inferiority of Traumed® gel compared to diclofenac gel
- to assess the tolerability and safety of Traumed<sup>®</sup> gel.

### Methodology:

Randomised, double-blind, active- and placebo-controlled confirmatory clinical trial.

### Number of Patients (Planned):

Estimation of sample size is based on the primary efficacy variable area under the curve (AUC) for pain on passive movement as measured by the Visual Analog Scale from baseline to Day 4. A two-sided test of equality of the study drug (Traumed® gel) and the comparator (placebo) at level 0.05 based on an expected raw scale treatment difference of AUC 25 [mm x days] and a common standard deviation of AUC 75 [mm x days] for the response variables (re-expressed for nonparametric evaluation in terms of the robust Mann-Whitney statistic as MW = 0.6), achieves a power of at least 90% for parametric first line analysis as well as for second line non-parametric analysis if the sample size is set to 291 patients for the Traumed® gel group and to 146 patients for the placebo group. Due to an additional safety requirement that AEs with incidence level of 1% for Traumed® gel are found during the study with probability 95%, 299 patients for the Traumed® gel group are required. Assuming a drop-out rate from the Safety Analysis Set of about 4% an amount of 312 randomized patients in the Traumed® gel group is needed. With an allocation ratio of 2:1:1 (Traumed® gel: diclofenac gel: placebo) we obtain 156 patients in the diclofenac and placebo group each, that is, a total of 624 patients with acute unilateral Grade 1 or Grade 2 sprain of the lateral ankle.

| Sponsor:<br>Biologische Heilmittel Heel<br>GmbH | Name of Medical Product:<br>Traumed® Gel | Active Ingredient(s): Homeopathic preparation, containing herbal and mineral ingredients as described in the Clinical Study Protocol |
|---|---|---|
| EudraCT number: 2016-004792-50 | | Indication: Acute ankle sprain |

In order to ensure the predefined power of the trial, a sample size enhancement is introduced for compensation of:

· cases for whom maintenance of blinding procedures may have been compromised.

For compensation, the final sample size will be enhanced to 202 patients for the diclofenac and Placebo group each, and to 404 patients for the Traumed® gel group resulting in a new total of 808 patients.

For more details see [protocol] sections 11.1.3 and 11.4. (revised per Amendment to protocol version 3.0)

### Diagnosis and Inclusion Criteria:

The patients have to meet all of the following inclusion criteria:

- 1. Acute unilateral Grade 1 or Grade 2 sprain of the lateral ankle
- 2. >18 years of age
- 3. Legally competent male or female outpatient
- 4. Injury occurred within previous 24 hours before first treatment expected
- Signed Informed Consent
- After 5 minutes of rest, pain on passive movement by investigator measured by Visual Analog Scale (VAS) >50 mm
- 7. Not pregnant (as proven by negative pregnancy test in case of woman of childbearing potential before first study drug administration) or breast-feeding. Females of childbearing potential must agree to maintain highly effective birth control throughout the study (see all details in [protocol] section 9.6). Such methods include:
  - oral, intravaginal, transdermal combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation,
  - oral, injectable, implantable hormonal contraception associated with inhibition of ovulation, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner (if received medical assessment of the surgical success), sexual abstinence (only if defined as refraining from heterosexual intercourse during the entire period of trial participation)

| <b>Sponsor:</b><br>Biologische Heilmittel Heel<br>GmbH | Name of Medical Product:<br>Traumed <sup>®</sup> Gel | Active Ingredient(s): Homeopathic preparation, containing herbal and mineral ingredients as described in the Clinical Study Protocol |
|---|---|---|
| EudraCT number: 2016-004792-50 | | Indication: Acute ankle sprain |

### **Exclusion Criteria:**

Potential study patients will be excluded if at least one of the following exclusion criteria is present:

- 1. Similar injury affecting the same joint within the past 6 months
- 2. Bilateral ankle injury
- 3. Grade 3 ankle sprain
- 4. Fracture of the ankle (It should be excluded by using e.g. the Ottawa Ankle Rules. In case of any doubt the exclusion of fracture by x-ray should be considered as per standard of care)
- 5. Chronic joint disorders such as clinically relevant osteoarthritis or aseptic arthritis
- 6. Disorders that may lead to joint oedema for other reasons than ankle sprain (such as heart failure, thrombosis, lymphedema and others)
- Diagnosis requiring bed rest, hospitalization, surgery, or use of any cast during the planned treatment period
- 8. Debilitating acute or chronic illness
- 9. Use of systemic and/or topical corticosteroids in the previous 8 weeks, any analgesics (e.g. paracetamol/ acetaminophen) in the previous 24 hours before Screening Visit, or 48 hours in the case of long-acting non-steroidal anti-inflammatory drug (NSAID), cyclooxygenase type 2 (COX-2) specific inhibitors, or tramadol and other opioids. Low dose acetylsalicylic acid (70 100 mg per day) for anti-thrombotic therapy is permitted if doses are stable for the month prior to Screening Visit and planned to be stable during the entire study
- History of sensitivity to any component of the study drugs (including e.g. paracetamol/ acetaminophen intolerance; patients in whom asthma attacks, skin rash or acute rhinitis are triggered by acetylsalicylic acid or non-steroidal anti-inflammatory drugs (NSAIDs)
- 11. Unwilling or unable to comply with all the requirements of the study protocol
- 12. Concurrent injury to proximal structures in ipsilateral lower extremity (i.e. concurrent shin, knee, thigh, or hip injury)
- 13. History of ligament avulsion, fracture or surgery to the affected lower extremity
- Presence of infections and/or skin diseases in the area of the study treatment site (including psoriasis)
- 15. Any previous treatments of the injured ankle, whether topical or systematic, are prohibited except RICE (simultaneous combination of all 4 elements Rest, Ice, Compression and Elevation which is restricted to be used until starting treatment with the investigational drug)
- 16. Participation in any clinical study within the past 4 weeks
- 17. Any relationship of dependence with the sponsor or with the investigator

### Test Product, Dose, and Mode of Administration:

Traumed<sup>®</sup> gel, 3 g of gel three times daily for 7 days, to sufficiently cover the area of the ankle, applied by gentle rubbing.

### Reference Product, Dose, and Mode of Administration:

Diclofenac 1% gel, 3 g of gel three times daily for 7 days, to sufficiently cover the area of the ankle, applied by gentle rubbing.

### Placebo therapy, Dose, and Mode of Administration:

Corresponding placebo gel formulation, 3 g of gel three times daily for 7 days, to sufficiently cover the area of the ankle, applied by gentle rubbing.

### Rescue medication, Dose and Mode of Administration:

Paracetamol (acetaminophen), 500 mg/tablet when necessary (pro re nata, PRN) for pain with a maximum of 4 tablets or 2000 mg/day (but not more than 2 tablets at a time), is permitted as rescue medication for relieving pain in all three treatment groups. Patients will not be allowed to take paracetamol within 8 hours prior to visit 2. For further visits the restriction is 24 hours. The intake will be recorded by the patients on the patient diary cards.

### Supportive therapy:

All patients receive soft support (elastic bandage) at Day 1. All patients will continue using soft support, however patients with Grade 2 will receive a semi-rigid removable brace after the evaluations at Day 7. These semi-rigid braces will be provided to all patients centrally and the investigator team will be trained for correct use at the investigator meeting to ensure standardized circumstances. In addition, using arm crutches will be strongly recommended at least until Day 4.

### Criteria for Evaluation:

### Primary Efficacy Variable

Area under the curve (AUC)\* for pain on passive movement in Visual Analog Scale (VAS) from baseline to Day 4

\*All AUC calculations will be based on actual time of measurement

### Secondary Efficacy Variables

- · AUC for pain at rest in VAS from baseline to Day 4
- AUC for pain on passive movement in VAS from baseline to Day 2, 7 and Final Visit
- AUC for pain at rest in VAS from baseline to Day 2, 7 and Final Visit
- Change from baseline of pain on passive movement in VAS to Day 4, 7 and Final Visit
- Change from baseline of pain at rest in VAS to Day 4, 7 and Final Visit
- Change from baseline to Day 2, 4, 7 and Final Visit in the Foot and Ankle Ability Measure (FAAM) Activities of Daily Living (ADL) subscale
- Amount of rescue medication (doses)
- Time to 50% improvement of pain at rest measured by VAS.

### Safety Variables

- Adverse Events (AEs)
- · Other observations related to safety (physical examinations and vital signs).

### Statistical Methods:

The summaries of the efficacy parameters, the statistical analyses of the primary efficacy variable, and the statistical analyses of the secondary efficacy variables will be performed on the Full Analysis Set (primary set for evaluation of superiority of Traumed® gel versus placebo, secondary set for evaluation of non-inferiority of Traumed® gel compared to diclofenac gel), and on the PP set (primary set for evaluation of evaluation of non-inferiority of Traumed® gel compared to diclofenac gel, secondary set for evaluation of superiority of Traumed® gel versus placebo).

Missing values for all efficacy parameters will be imputed by the last observation carried forward (LOCF) approach. In addition, a last percentile carried forward approach (LPCF) will be performed as sensitivity analysis (see also [protocol] section 11.1.4). Further sensitivity analyses resulting from the blind review of the data will be provided in the final Statistical Analysis Plan.

All statistical tests will be two-sided with a significance level of  $\alpha$ =0.05, unless specified otherwise. Where appropriate, statistical tests will be supported by presenting estimates and 95% confidence intervals for the respective treatment effects and differences between the treatment groups. These estimates and confidence intervals will be based on the respective statistical models used for the analysis.

### Confirmatory analyses

- AUC for pain on passive movement in VAS from baseline to Day 4 (test for superiority, Traumed® gel versus placebo), Full Analysis Set (FAS)
- AUC for pain on passive movement in VAS from baseline to Day 4 (test for non-inferiority, Traumed® gel versus diclofenac gel), Per-Protocol Analysis Set (PP)

If the first *a priori* ordered test (superiority) shows statistical significance, the subsequent hypothesis (non-inferiority) can then be tested individually in a confirmatory manner according to the principle of *a priori* ordered hypotheses (for control of alpha using stepwise testing see [Maurer et al. 1995]).

Clinical safety will be addressed by assessing AEs, physical examinations, vital signs and as needed laboratory assessments in a descriptive manner.

| Contract Research Organisation: | AMS Advanced Medical Services GmbH |
|---------------------------------|------------------------------------|
| | Am Exerzierplatz 2 |
| | D-68167 Mannheim |
| | Phone: +49 621 700 95 100 |
| | Fax: +49 621 700 95 140 |
| Statistician: | idv Datenanalyse & Versuchsplanung |
| | Tassilostrasse 6 |
| | D-82131 Gauting/ Germany |

# 6.2 Schedule of Study Procedures

| | Initial Visit<br>Screening/Baseline | Treatm<br>Visit 2 | ent Visits<br>Visit 3 | EoT Visit<br>Visit 4 | Final Visit<br>Visit 5 |
|---|---|---|---|---|---|
| | Day 1 | Day 2 | Day 4<br>+ 1 day | Day 7 | Day 14<br>+/- 1 day |
| Informed Consent | X | | , a only | | ,, 1 day |
| Inclusion/Exclusion Criteria | X | 2 | | | |
| Demographics | X | | | | |
| Pregnancy test (if applicable) | X | | | X | |
| Medical history | X | | | 25.5 | |
| Time and grading of injury | X | | * | | |
| Height/Weight (BMI) <sup>1</sup> | X | | | | X <sup>1</sup> |
| Physical examination including | | | | | |
| blood pressure and pulse | X | | | | X |
| Randomization | X | | | | |
| Dispense patient diary <sup>2</sup> | X | | X | | |
| FAAM-ADL <sup>3</sup> | X | X | X | X | X |
| Pain at rest by Visual Analog<br>Scale (VAS) <sup>3</sup> | Х | X | X | X | X |
| Pain on passive movement by<br>Visual Analog Scale (VAS) <sup>3</sup> | X | X | x | X | X |
| IMP tubes dispensed | X | | | | |
| Investigational treatment | X | X | X | X | |
| Application of soft support<br>(elastic bandage) | X | X | X | X | X<br>(as required) |
| Rescue medication dispensed | х | 2 | X<br>(if needed) | (as required) X (if needed) | (us requires) |
| Diary reviewed | | X | X | X | X |
| Diary returned | | | X | | X |
| IMP tubes weighted | | | X | X | |
| Rescue medication reviewed | | X | X | X | X |
| IMP tubes returned and sealed | | Λ | A | X | - A |
| Rescue medication returned | * | | * | 24 | X |
| Check use of other pain<br>medication and record if any | X | X | X | X | X |
| Record previous/concomitant medication | х | X | Х | х | X |
| Record Adverse Events <sup>4</sup> | v | v | 222 | v | 200 |
| Record use of arm crutches | X | X | X<br>X | X<br>X | X |
| Confirmatory check of grading | Λ | Λ | X | Λ | Α |
| Application of semi-rigid brace<br>for Grade 2 | | S | Λ | X | X |
| Question to patients which<br>treatment they assume to have<br>received | | 5 | 3 | | Х |

<sup>&</sup>lt;sup>1</sup> At Visit 5 (day 14) only the weight will be measured.

<sup>2</sup> The first patient diary will be collected on Day 4. The patient will receive second diary on the same day.

<sup>3</sup> The time point of each visits/measurements of patients shall be ideally the same at each visit (+/- 1 hour). 4 Including adverse events observed at the site of administration of the IMP (lateral ankle).

## 6.3 Assessment of Efficacy

### 6.3.1 Primary Efficacy Parameter

Pain assessment on VAS for evaluating pain on passive movement

Ankle pain will be measured using a 100 mm VAS starting with no pain (0 mm) and ending with most severe imaginable pain the patient may imagine in relation to his/her ankle sprain (100 mm).

First the patients will be asked after 5 minutes rest to assess their pain themselves on a VAS scale for a secondary efficacy assessment (for details see [protocol] section 6.3.2).

Than while the patient is still at rest the investigator should perform 10° dorsal- and 30° plantar flexion on the injured ankle and the patients will assess their pain themselves on a VAS scale (primary efficacy assessment). The range of movement will be controlled by using a goniometer. It is very important that no lateral move of the ankle joint will be made. The pain to be assessed is the pain on passive movement.

To ensure a consistent assessment between investigators, investigators will be trained together at the investigator meeting.

The date and time of assessment will be recorded. Pain assessments should take place +/- 1 hour related to baseline at each visit for the individual patient, whenever possible.

### 6.3.2 Secondary Efficacy Parameters

Pain assessment on VAS for evaluating pain at rest

Ankle pain will be measured using a 100 mm VAS starting with no pain (0 mm) and ending with most severe imaginable pain the patient may imagine in relation to his/her ankle sprain (100 mm).

The patients will be asked after 5 minutes rest to assess their pain themselves on a VAS scale.

Foot and Ankle Ability Measure (FAAM), Activities of Daily Living (ADL)

The FAAM is a validated questionnaire and was developed to meet the need for a self-reported evaluative instrument that comprehensively assesses physical function of individuals with musculoskeletal disorders of the leg, foot, and ankle.

It is a well-established and widely used responsive multidimensional outcome measure with a sensitivity capable of detecting subject-relevant symptoms and clinically significant changes in health in ankle sprain.

The FAAM-ADL/S consists of an ADL (21-item scale) and a sports (S) subscale (8 items) asking study participants to rate their ability to perform specific tasks. The FAAM-ADL/S is a valid and reliable instrument in the public domain (Martin 2005, Carcia et al. 2008).

The possible responses for each item are the following: no difficulty, slight difficulty, moderate difficulty, extreme difficulty, unable to do and not applicable.

In this clinical trial FAAM-ADL will be used. The scoring of the FAAM-ADL will be performed according to the recommendations of Martin et al. 2005.

The response to each item on the FAAM-ADL subscale will be recorded from 4 to 0, with 4 being 'no difficulty' and 0 being 'unable to do'. Responses marked as not applicable will not counted. The scores on each of the items will be added together to get the item score total. The total number of items with a response is multiplied by 4 will get the highest potential score. If all 21 items are answered, the highest potential score will be 84. If one item is not answered the highest potential score will be 80, if two are unanswered the highest potential score will be 76. The total item score will be divided by the highest potential score and then multiplied by 100 to produce the FAAM-ADL score that ranges from 0 to 100. According to the above recommendations the final scores of the FAAM-ADL subscale is to be standardized to a 0 - 100 scale (0 = worst score, 100 = best score).

# Time to 50 % improvement of pain measured by VAS

The time to 50 % improvement will be calculated from VAS assessments on pain at rest performed at all patient visits using the percent changes from baseline (recorded at Day 1).

### Rescue medication

The rescue medication use will be documented in the eCRF based on the information given in the patient diary and the drug accountability for rescue medication during the study.

## 6.3.3 Safety Assessments

In this study topical medications are applied for a local disorder where systemic effects are neither expected from the disorder nor from any of the investigational medications given. Due to these reasons, no safety laboratory testing is planned for this study.

### **Adverse Events**

Definition, collection and reporting of adverse events are described in [protocol] section 9.

### Vital Signs

Vital signs (heart rate, systolic/ diastolic blood pressure) will be collected and evaluated by comparison of the results obtained pre- and post-treatment.

### Physical examination

At screening/ baseline and at final visit a physical examination will be performed. Physical status of cardiovascular, respiratory musculoskeletal and gastrointestinal systems, head and eyes and in addition other abnormalities if applicable will be recorded in the eCRF.

Any clinically significant change observed at the final evaluation of vital signs and physical examination in comparison with baseline has to be evaluated carefully, recorded as AE if abnormal, and a possible causality will be evaluated (see [protocol] section 9.3.2).

### 7. BLIND DATA TRANSFERS AND QUALITY ASSURANCE

The blind data transfers from the CRO responsible for the eCRF (AMS Advanced Medical Services GmbH) to IDV was performed according to the IDV Data Transfer Guideline Version Final 1.0 from 13 December 2017.

The following data transfers were performed for risk-based centralized statistical monitoring:

- INTERIM TRANSFER:
  - 1. 28.05.2018 (TRAUMED-2018-05-28 01)
  - 2. 26.06.2018 (TRAUMED-2018-06-26 02)
  - 3. 03.09.2018 (TRAUMED-2018-09-03 03)
  - 4. 08.11.2018 (TRAUMED-2018-11-08 04)
  - 5. 15.01.2019 (TRAUMED-2019-01-15 05)
  - 6. 11.03.2019 (TRAUMED-2019-03-11 06)
  - 7. 12.04.2019 (TRAUMED-2019-04-12 07)
  - 8. 13.05.2019 (TRAUMED-2019-05-13 08)
  - 9. 09.09.2019 (TRAUMED-2019-09-09 09)
  - 10. 18.11.2019 (TRAUMED-2019-11-18\_10)
  - 11. 14.01.2020 (TRAUMED-2020-01-14 11)
  - 12. 11.07.2020 (TRAUMED-2020-07-11 12)
  - 13. 11.09.2020 (TRAUMED-2020-09-11 13)
  - 14. 10.11.2020 (TRAUMED-2020-11-10 14)
  - 15. 02.12.2020 (TRAUMED-2020-12-02 15)
- SOFTLOCK TRANSFER:
  - o 18.01.2021 (TRAUMED-2021-01-18 16)
  - o 20210113 C1502 Issue Overview FINAL
- HARDLOCK TRANSFER:
  - o 29.03.2021 (TRAUMED-2021-03-29 17)

Based on the hardlock data, patients with major protocol deviations are coded on the base of the definitions in the final Statistical Analysis Plan. The major protocol deviations leading to exclusion from analysis sets as well as the final datasets (analysis populations) are documented on a per patient base in the Appendix of the final Statistical Analysis Plan.

### 8. CHANGES TO THE PROTOCOL

# Preliminary Remark on Substantial Protocol Amendment version 4.0 (February 3, 2020) to Protocol version 3.0

A total of 184 'issue patients', for whom maintenance of blinding procedures may have been compromised, have been identified in 2019 after re-examination of adherence to blinding specifications by the local monitors. Rationale for the re-examination were corresponding findings from site inspections by the German Local Authorities in 2019 (Gesundheitsamt Düsseldorf of German Federal State North Rhine Westphalia, NRW). Re-training and close follow-up control for the sites was implemented to prevent occurrence of further issue cases.

In order to ensure the pre-defined power of the trial for the trial objectives, including the confirmatory test for non-inferiority (Traumed® gel compared to diclofenac gel) based on the Per-Protocol Analysis Set (PP), a sample size enhancement was introduced by means of Protocol Amendment version 4.0 to Protocol version 3.0 for compensation of cases for whom maintenance of blinding procedures may have been compromised.

As specified in C1502 Study Protocol Version 4.0 (3 February 2020) and in the Amendment Summary Document for Substantial protocol Changes (3 February 2020), detailed handling of these problem cases have to be defined in this update of the Statistical Analysis Plan (SAP).

Based on the Blind Data Review Meeting from March 09, 2021 (C1502\_MTG\_NOTES\_BDRM\_09MAR2021\_20210324), the operational handling as specified in the following section shall ensure the integrity and validity of the trial.

### OLD

(Final C1502 Study Protocol Version 4.0, Amendment to Protocol version 3.0)

In order to ensure the data integrity of the trial and to exclude potential bias introduced by partial unblinding, a separate analysis of problematic and non-problematic cases will be conducted with subsequent meta-analytic pooling and test for overall effect and heterogeneity.

Further details will be defined in an update of the Statistical Analysis Plan (SAP).

## NEW

(Final BDRM decision)

In order to ensure the data integrity of the trial and to exclude potential bias introduced by partial unblinding, a separate analysis of problematic and non-problematic cases will be conducted. All confirmatory and secondary analyses will be based on the group of non-issue patients. Results of issue patients will be provided separately in the Appendix of the Clinical Trial Report (CTR).

### RATIONALE

Blind data review revealed severe deviations of 'issue' cases from 'non-issue' cases, suggesting that compromised cases might constitute a serious risk of bias, preventing pooled analysis.

The multivariate P-values for the comparison of issue cases vs. non-issue cases regarding the three key domains "Baseline", Efficacy", and "RICE", were throughout below 0.0001, thus, suggesting serious structural differences between issue cases and non-issue cases. The rate of <u>major</u> protocol violations was significantly higher in the group of issue cases (11.4%) as compared to non-issue cases (1.9%; P<0.0001). Also the patient's guess on which treatment he/she received was less balanced in the issue group as compared to the non-issue group (patient's guess for the two <u>active</u> treatments: non-issue cases: 39% Traumed vs. 35% diclofenac, issue cases: 42% Traumed vs. 29% diclofenac).

Final BDRM Decision: In order to preserve the integrity and validity of the trial, issue patients will not be included into the pre-planned confirmatory and secondary analyses of the main part of the Clinical Trial Report. While being evaluated for baseline characteristics, efficacy and safety endpoints in the same way as the non-compromised cases, the compromised cases will be reported separately in the Appendix of the Clinical Trial Report (results to be interpreted with care due to the described issues).

As stated before, the sample size was already proactively increased for compensation in case of an exclusion of the issue patients (Protocol Amendment version 4.0 from February 3, 2020 to Protocol version 3.0). The Reason/Justification for Change of Protocol Section 11.4 (Protocol Amendment version 4.0 from February 3, 2020 to protocol version 3.0) was provided in the Amendment Summary Document for Substantial Protocol Changes (SOC document from February 3, 2020):

The enhancement will ensure planned power and validity for evaluating the pre-defined trial objectives also in case that **only non-compromised cases** allow valid and unbiased conclusions ...

# 9. ADDITIONAL SPECIFICATIONS TO THE PROTOCOL

# 9.1 Standard Procedures

Within the framework of the idv system, the following standard ensemble of classic and
robust summarizing statistics will be provided for data description: mean, standard
deviation, standard error of the mean, minimum, lower quartile, median, upper quartile,
maximum, valid number. In addition, measures for skewness and kurtosis will be
provided for suitable efficacy variables. Where appropriate, the result presentation will
include changes from baseline.

• For categorical data, frequency counts will be provided with their associated percentages. Semi-quantitative and quantitative efficacy data will be additionally visualized by boxplot diagrams. All standardized effect sizes (Mann-Whitney) will be visualized with their corresponding 95%-confidence intervals. All standard statistical tables are generated with the standard table layout of the validated statistical package TESTIMATE V6.5.14 (IDV Gauting). Associated meta-data and variable labels are finalized before unblinding. All standard scientific figures are generated with the standard figure layout of the validated scientific package SCIENCEGRAPH V4.9.39 (IDV Gauting).

# 9.2 Demography and Baseline Characteristics

### 9.2.1 Operationalizations in Final Protocol

None.

### 9.2.2 Additional Operationalizations

- Besides standard descriptive analyses (see section 9.1), formal homogeneity analyses for demographic variables and baseline characteristics will be performed based on the full analysis set (FAS) and the per-protocol set (PP). Robust Mann-Whitney estimators and their 95% confidence intervals will used as standardized summary measures across the relevant demographic-anamnestic variables (demography, physical examination, vital signs, supportive therapy, time and grading of injury) as well as across the efficacy criteria at baseline (VAS pain on passive movement, VAS pain at rest, FAAM). This will be performed in order to check baseline comparability of the three randomized groups in a robust, nonparametric way (minimized assumptions, independent from data type).
- As benchmark for relevant baseline differences, a Mann-Whitney estimator of 0.36 and 0.64 respectively will be applied (referring to a standardized difference of 0.5 according to Cohen, which is regarded as a medium-sized difference).
- In the case of inhomogeneities, stratified analyses will be performed by means of the Peto-Wilcoxon test (2 sided; 95% confidence interval, CI) with adjustment within the framework of the Cochran-Mantel-Haenszel pooling procedure (CMH pooling, also known as van Elteren pooling). For this purpose, depending on the respective data type and distribution, nominal categories, medians or quartiles of the affected baseline criteria will be used for stratification.

# 9.3 Evaluations and Endpoints – First Line Analysis

# 9.3.1 Primary Efficacy Variable

# 9.3.1.1 Operationalizations in Final Protocol

## **Primary Efficacy Variable**

Area under the curve (AUC)\* for pain on passive movement in Visual Analog Scale (VAS) from baseline to Day 4

# **Confirmatory Analyses**

1. AUC for pain on passive movement in VAS from baseline to Day 4 (test for superiority, Traumed<sup>®</sup> gel versus placebo), Full Analysis Set. The null and alternative hypotheses for the comparison of Traumed<sup>®</sup> gel versus placebo can be formulated as follows:

H<sub>0</sub>:  $\mu_T = \mu_P$ H<sub>A</sub>:  $\mu_T \neq \mu_P$ 

H<sub>0</sub>: Null hypothesis; H<sub>A</sub>: Alternative Hypothesis; T: Test Treatment; P: Placebo Treatment; μ: mean of population (AUC)

2. AUC for pain on passive movement in VAS from baseline to Day 4 (test for non-inferiority, Traumed® gel compared to diclofenac gel), Per-Protocol Analysis Set (PP). For the comparison of Traumed® gel versus diclofenac gel the null and alternative hypothesis can be formulated as follows:

H<sub>0</sub>:  $\mu_{T} - \mu_{R} > 25 \text{ [mm x days]}$ 

H<sub>A</sub>:  $\mu_{\text{T}} \cdot \mu_{\text{R}} \leq 25 \text{ [mm x days]}$ 

 $H_0$ : Null hypothesis;  $H_A$ : Alternative Hypothesis; T: Test Treatment; R: Reference Treatment;  $\mu$ : mean of population (AUC)

Hypothesis no. 1 (superiority) is based on the FAS analysis set, while hypothesis no. 2 (non-inferiority) is based on the PP analysis set. This way, both hypotheses are based on the more conservative data set.

If the first *a priori* ordered test (superiority) shows statistical significance, the subsequent hypothesis (non-inferiority) can then be tested individually in a confirmatory manner according to the principle of *a priori* ordered hypotheses (for control of alpha using stepwise testing see [Maurer et al. 1995]).

<sup>\*</sup>All AUC calculations will be based on actual time of measurement.

The confirmatory analyses will be performed using an analysis of covariance (ANCOVA) with baseline pain VAS as covariate. Due to the expected small number of patients per center, an additional inclusion of center as covariate will not be performed (see also EMA Guideline on adjustment for baseline covariates, section 4.2.3., EMA/295050/2013).

# 9.3.1.2 Additional Operationalizations

- Visit 4 (Day 7) will be introduced as additional primary endpoint in the chain of a priori ordered hypotheses, leading to the following final sequence of confirmatory analyses:
  - 1. AUC for pain on passive movement in VAS from baseline to Day 4 (test for superiority, Traumed® gel versus placebo)
  - 2. AUC for pain on passive movement in VAS from baseline to Day 4 (test for non-inferiority, Traumed® gel compared to diclofenac gel)
  - 3. AUC for pain on passive movement in VAS from baseline to Day 7 (test for superiority, Traumed® gel versus placebo)
  - 4. AUC for pain on passive movement in VAS from baseline to Day 7 (test for non-inferiority, Traumed® gel compared to diclofenac gel)

If the preceding *a priori* ordered test shows statistical significance, the subsequent hypothesis can then be tested individually in a confirmatory manner according to the principle of *a priori* ordered hypotheses (for control of alpha using stepwise testing see [Maurer et al. 1995]).

**Comment:** The original endpoints at Day 4 remain unchanged (hypotheses no. 1 and no. 2), however Day 7 is introduced as additional primary endpoint in the chain of *a priori* ordered hypotheses (hypotheses no. 3 and no. 4). This addition is implemented as per BDRM decision in order to avoid lack of assay sensitivity at the early stage of the ankle joint injury (C1502\_MTG\_NOTES\_BDRM\_09MAR2021\_20210324).

- Descriptive procedures will be performed according to section 9.1.
- For the analysis of covariance, in addition to the table with descriptive statistics and the
  analysis of variance of the covariate (test for homogeneity of the groups with respect to
  the covariate), the following results of the analysis of covariance will be generated:
  - Analysis of covariance of the full model (separate regression lines for each group) with the following information:
    - Test for parallelism and group difference at X<sub>0</sub> as an indication of group differences in case the regression lines are not parallel (for the hypothesis of parallelism a 10%-level will be applied).

- Model parameter: for each group, the point of intersection of the regression line, the slope and the adjusted mean value of X<sub>0</sub>, the common mean value of the covariates for all groups.
- Analysis of covariance for the reduced regression model (a single regression line for all groups for the assumption that the regression lines are parallel), with the following information:
  - Covariates (within), an indication of the significance and relevance of the covariate for the criterion.
  - Test statistic for adjusted group differences, correct also for groups of unbalanced size.
  - Coefficient of determination R<sup>2</sup> for the amount of variation of the criterion, which is explained by the covariate and the differences between the groups.
  - Model parameter: the y-intercept and slope of the regression lines (slopes are now necessarily identical because of the reduction of the full model), adjusted mean values for a common value X<sub>0</sub> of the covariate.
- The analysis of covariance of the full model will be used for the confirmatory approach (the reduced regression model is provided as supportive information only)
- Descriptive Procedures: TESTIMATE V6.5.14; PROC BASIC STATISTICS / SCIENCEGRAPH V4.9.39
- Test Procedures: TESTIMATE V6.5.14; PROC ANALYSIS OF COVARIANCE

# 9.3.2 Secondary Efficacy Variables

# 9.3.2.1 Operationalizations in Final Protocol

# Secondary Efficacy Variables

- AUC for pain at rest in VAS from baseline to Day 4
- AUC for pain on passive movement in VAS from baseline to Day 2, 7 and Final Visit
- AUC for pain at rest in VAS from baseline to Day 2, 7 and Final Visit
- Change from baseline of pain on passive movement in VAS to Day 4, 7 and Final Visit
- Change from baseline of pain at rest in VAS to Day 4, 7 and Final Visit
- Change from baseline to Day 2, 4, 7 and Final Visit in the FAAM-ADL subscale
- Amount of rescue medication (doses)
- Time to 50% improvement of pain at rest measured by VAS at patient visits.

# 9.3.2.2 Additional Operationalizations

- AUC for pain on passive movement in VAS from baseline to Day 7 is defined as additional primary endpoint (see section 9.3.1.2), and, thus, removed from secondary efficacy variables.
- Descriptive procedures for secondary efficacy variables (1) to (7) will be performed according to section 9.1. Descriptive procedures for secondary efficacy variable 'time to 50% improvement' will be performed by means of frequency counts based on patient visits (50% improvement of pain at rest), as well as by Kaplan-Meier curves for time-to-event (including censored values). In addition to pain at rest (measured by VAS at patient visits), also pain on passive movement will be evaluated applying the same procedures.
- Test procedures for secondary efficacy variables (1) to (6) will be performed for the FAS and PP analysis sets as specified for the primary efficacy variable by analysis of covariance (see section 9.3.1.2), applying the associated baseline pain VAS as covariate. The test procedure for the secondary efficacy variable (7) will be performed for the FAS and PP analysis sets as specified for the primary efficacy variable by analysis of covariance (see section 9.3.1.2), applying baseline pain on passive movement in VAS as covariate. The secondary efficacy variable (8) will be analyzed by means of the Peto-Logrank test (time-to-event (logrank) test).
- Descriptive Procedures (Secondary Efficacy Variables (1) to (7)): TESTIMATE V6.5.14; PROC BASIC STATISTICS / SCIENCEGRAPH V4.9.39

- Descriptive Procedures (Secondary Efficacy Variable (8)): TESTIMATE V6.5.14;
   PROC KAPLAN-MEIER FUNCTION / SCIENCEGRAPH V4.9.39
- Test Procedures (Secondary Efficacy Variables (1) to (7): TESTIMATE V6.5.14;
   PROC ANALYSIS OF COVARIANCE
- Test Procedures (Secondary Efficacy Variable (8): TESTIMATE V6.5.14; PROC PETO-LOGRANK-TEST

## 9.4 Evaluations and Endpoints – Second Line Analysis

### 9.4.1 Nonparametric Analysis

## 9.4.1.1 Operationalizations in Final Protocol

As a sensitivity analysis to the primary parametric approach, a nonparametric analysis will be performed for the two primary hypotheses.

The nonparametric procedures will be performed by means of the Wilcoxon-Mann-Whitney test. The Wilcoxon-Mann-Whitney test (WMW test) is the well-known robust test attributed to Wilcoxon (Wilcoxon 1945) and Mann and Whitney (Mann et al. 1947); for details of the test see e. g. Armitage, Berry, and Matthews (Armitage et al. 2002), or Sprent and Smeeton (Sprent et al. 2001).

The Mann-Whitney estimator (MW) is the associated effect size measure for the Wilcoxon-Mann-Whitney test (WMW test). It is a robust but highly sensitive effect size measure to determine the magnitude and direction of the treatment effects. It is recommended by many authors for its sensitivity and robustness in all data situations (Agresti et al. 1984, Brunner et al. 2000, Munzel et al. 2003, D'Agostino et al. 2006, Brunner et al. 2013, Kieser et al. 2013) for ordinal scales in non-inferiority trials it is even regarded as the 'gold standard' see, e.g. Design and Analysis of Non-Inferiority Trials (Rothmanns et al. 2011). Technically, the MW gives the probability that a randomly chosen subject of the test group is better off than a randomly chosen subject of the comparison group (with the probability ranging from 0 to 1, with 0.5 indicating equality); it is statistically defined as: P (X<Y) + 0.5 P (X=Y).

The relevant benchmarks for the Mann-Whitney effect size measure (MW) are as follows (Colditz et al. 1988):

| 0.29 | large inferiority |
|------|--------------------------|
| 0.36 | medium sized inferiority |
| 0.44 | small inferiority |
| 0.50 | equality |
| 0.56 | small superiority |
| 0.64 | medium sized superiority |
| 0.71 | large superiority |

Under the assumption of a normal distribution the defined non-inferiority margin AUC 25 mm x days with common standard deviation 75 mm x days, (see [protocol] section 11.4) can be re-expressed in terms of the Mann-Whitney statistic: the raw scale margin results in a standardized mean difference of 25/75 = 0.33, which can be directly transformed to a Mann-Whitney margin of 0.407 (Rahlfs et al. 2014). This margin is consistent with the nonparametric NI bound of 0.40 in a previous NI trial (Gonzalez et al. 2013).

In addition, a non-parametric repeated measurement analysis will be performed by means of the generalized Wilcoxon-Mann-Whitney test (Wei-Lachin procedure), combining the repeated observations by a simultaneous, directional test.

# 9.4.1.2 Additional Operationalizations

- The nonparametric procedures will be performed for the FAS and PP analysis set as sensitivity analyses for the primary parametric approach. The univariate analysis will be performed by means of the Wilcoxon-Mann-Whitney (WMW) test for the area under the curve (AUC) of pain on passive movement in Visual Analog Scale (VAS) from baseline to Day 4. The repeated measurement analyses will combine the repeated observations of pain on passive movement (VAS) at Day 2, 4, 7 and Final Visit by means of the generalised Wilcoxon-Mann-Whitney test (Wei-Lachin procedure, directional test).
- Descriptive Procedures: TESTIMATE V6.5.14; PROC BASIC STATISTICS / SCIENCEGRAPH V4.9.39
- Test Procedures: TESTIMATE V6.5.14; PROC WILCOXON-MANN-WHITNEY-U-TEST / SCIENCEGRAPH V4.9.39 / PROC MULTIVARIATE COMPARISONS -WEI-LACHIN – DIRECTIONAL

### 9.4.2 Stratification

# 9.4.2.1 Operationalizations in Final Protocol

In order to control for center effects, a robust stratified analysis will be performed for the primary efficacy criterion applying the Cochran-Mantel-Haenszel procedure with adjustment for centers (CMH pooling, also known as van Elteren pooling). This procedure is robust also with very low sample sizes per center and group.

In order to control for effects of delayed "Day 4" assessments (Day 4+1), a robust stratified analysis (CMH) will be performed for patients with and without delay.

In order to ensure the data integrity of the trial and to exclude potential bias introduced by partial unblinding, a separate analysis of problematic and non-problematic cases will be conducted with subsequent meta-analytic pooling and test for overall effect and heterogeneity.

Further details will be defined in an update of the Statistical Analysis Plan (SAP). (revised per Amendment to protocol version 3.0)

# 9.4.2.2 Additional Operationalizations

- The robust stratified analyses will be performed for the FAS and PP analysis set as sensitivity analyses for the primary parametric approach by means of the Cochran-Mantel-Haenszel (CMH) pooling procedure with Wilcoxon scores (Peto-Wilcoxon test).
  - Adjustment for centers by means of the CMH pooling procedure will be performed for the area under the curve (AUC) of pain on passive movement in Visual Analog Scale (VAS) from baseline to Day 4 with centers as strata. Small centers will technically be pooled. According to protocol, the final pooling benchmark is to be decided at the time of the blind review of the soft lock data with documentation in the final Statistical Analysis Plan (see ICH Guidance E9 §3.2 "any case decisions concerning this approach should always be taken blind to treatment, for example at the time of the blind review"). Based on the softlock data, the pooling benchmark for small centers is set to N<20 (virtual center labelled as "center 99"). This way, the sensitivity analysis will be based on 12 center strata and one virtual center, which is regarded as reasonable procedural size for the sensitivity analysis.</p>
  - Adjustment for patients with and without delayed "Day 4" assessments (Day 4+1) will be performed for the area under the curve (AUC) of pain on passive movement in Visual Analog Scale (VAS) from baseline to Day 4.
- Due to serious risk of bias, the "problematic" cases will be evaluated separately and will not be part of the confirmatory or secondary analyses (for details, see section 8 Changes to the Protocol).
- Test Procedures: TESTIMATE V6.5.14; PROC PETO-WILCOXON-TEST.

## 9.5 Accounting for Missing Data

# 9.5.1.1 Operationalizations in Final Protocol

The pre-planned analysis procedures are as follows:

# 1. Last Observation Carried Forward [LOCF] (Applied to all Efficacy Analyses)

A LOCF analysis (Last Observation Carried Forward) will be performed as first line analysis. LOCF will be applied for missing values regardless of the reason for discontinuation.

# 2. Last Percentile Carried Forward [LPCF] (Applied as Sensitivity Analysis to the First Line Efficacy Analyses)

The LPCF method carries forward the change information, using the percentile value with back transformation to raw scale, instead of last value carried forward. This approach was recently developed and recommended by O'Brien, Zhang and Bailey in 2005 (O'Brien et al. 2005). The results of this method are well comparable to the mixed-effect models for repeated measures (MMRM), without making the corresponding parametric assumptions. According to their simulation study the calculated estimators should be negligibly biased by missing data.

Additional sensitivity analyses resulting from the blind review of the data and further technical details will be provided in this final Statistical Analysis Plan.

The frequency and type of missing values will be documented in the Clinical Trial Report.

## 9.5.1.2 Additional Operationalizations

- The imputation by means of Last Observation Carried Forward [LOCF] will be applied to all first line analyses (confirmatory and exploratory) with the exception of the secondary efficacy variables no. 7 and 8 (see section 9.3.2). Imputation of missing values is performed using the last existing follow-up value. The imputation by means of Last Percentile Carried Forward [LPCF] will be omitted due to the marginal number of missing efficacy values.
- The number of non-missing values will be documented in the Clinical Trial Report for all variables and evaluations (valid number). The frequency and type of missing values will be documented in the Clinical Trial Report for the primary efficacy variable (area under the curve, AUC) of pain on passive movement in Visual Analog Scale (VAS) from baseline to Day 4.
- The standard ensemble of classic and robust summarizing statistics (see section 9.1) will be provided for the pre-specified imputation as well as for *data as available*, i.e. without imputation.

# 9.6 Evaluations and Endpoints – Safety

# 9.6.1.1 Operationalizations in Final Protocol

### Safety variables are:

- AEs
- other observations related to safety (physical examinations, vital signs).

All safety summaries will be performed on the Safety Analysis Set if not indicated otherwise. For vital signs, no formal testing will be applied to detect imbalances between the treatment groups.

AEs will be presented by MedDRA Preferred Term and System Organ Class in different categories.

Incidence rates of AEs, SAEs and AEs related to investigational product will be reported. The duration of exposure to IMP and the amount of IMP used for the three treatment groups (Traumed® gel, diclofenac gel and placebo gel) will be analyzed.

# 9.6.1.2 Additional Operationalizations

Descriptive procedures will be performed according to section 9.1.

## 9.7 Analysis Populations

### 9.7.1.1 Operationalizations in Final Protocol

**Safety Analysis Set**: Randomized patients who receive at least one dose of investigational medication will form the Safety Analysis Set. The Safety Analysis Set will be used for all analyses of safety, tolerability, and background characteristics. For this set, the exposure to IMP will be also analysed.

**Full Analysis Set (FAS):** The Full Analysis Set is a subset of the Safety Analysis Set consisting of all patients with acute unilateral Grade 1 or Grade 2 sprain of the lateral ankle, for whom both baseline and Day 4 VAS values of pain are available. The Full Analysis Set will be used for the Intent-to-Treat (ITT) analysis.

**Per-Protocol (PP) Set:** Patients in the Full Analysis Set without major protocol deviations will form the PP Set. The PP Set will be used for the per-protocol analysis of the efficacy parameters. The same efficacy evaluations as in the FAS are planned. Relevant differences between the FAS and PPS will be evaluated in the Clinical Trial Report.
Protocol deviations will be collected during the entire trial and will be classified as minor or major at the Blind Data Review Meeting (BDRM). Protocol deviations that may affect the efficacy outcome of participants will be classified as major. The decision about major protocol deviations and assignments to populations will be documented in the BDRM minutes.

### 9.7.1.2 Additional Operationalizations

- In order to preserve validity and integrity of the trial, all confirmatory and secondary analyses will be based on the group of non-issue patients (for details see section 8 Changes to the Protocol). As stated in the 'Amendment Summary Document for Substantial Protocol Changes', the sample size was proactively enhanced to ensure planned power and validity for evaluating the pre-defined trial objectives also in case that only non-compromised cases allow valid and unbiased conclusions. Results of issue patients will be provided separately in the Appendix of the Clinical Trial Report (CTR).
- FAS: VAS availability at Day 4 is referring to LOCF (primary analysis).
- PP: premature discontinuations due to "lack of efficacy", "adverse event", or
  "lack of efficacy" and "adverse event" (i.e. drug-related premature
  discontinuations) will not be excluded from the PP analysis, regardless of any
  existing protocol deviation. Benchmarks for "Major Protocol Deviation" (final
  BDRM decisions):
  - Grade 3 determination after Visit 3
  - VASPM V1 < 50</li>
  - Missing VASPM at V1 or V3 (Related to ,Data as Available')
  - Visit 2 \leftrightarrow Day 2 (Protocol Day 2)
  - Visit 3 < Day 4 or > Day 5 (Protocol Day 4 + 1 Day)
  - Visit  $4 < \text{Day } 6 \text{ or } > \text{Day } 9 \text{ (Protocol Day } 7 \pm 1 \text{ day)}$
  - Compliance < 80% at V3 or V4
  - Premature Discontinuation (not drug-related)
  - The analysis populations (Safety, FAS, and PP) are listed individually in the Appendix of the final Statistical Analysis Plan.

#### 10. SOFTWARE APPLIED

Unblinded clinical trial evaluation will be performed on high security PCs (HSPC) within a validated working environment at the department 'Clinical Research/Biometry' in the institute IDV Data Analysis and Study Planning under supervision of Volker W. Rahlfs, PhD., C. Stat. (RSS), with a 'Certificate Biometry in Medicine GMDS'.

Software packages to be used for unblinded analyses and generation of Clinical Trial Report (CTR):

- TESTIMATE V6.5.14 (statistical analyses)
- SCIENCEGRAPH V4.9.39 (scientific figures)
- ICH-Study-Report-Manager V2.4.3 (Clinical Trial Report)

## 11. POST HOC CHANGES TO PLANNED ANALYSES (POST UNBLINDING)

Any major changes to this plan after final sign-off will be specified in the Clinical Trial Report of the final analyses with corresponding scientific rationales.

### 12. REFERENCES

- AGRESTI, A. 1984. Analysis of Ordinal Categorical Data, New York, NY, Wiley & Sons.
- ARMITAGE, P., BERY, G. & MATTHEWS, J. N. S. 2002. Statistical Methods in Medical Research, Malden, MA, Blackwell Science.
- ARORA, S., HARRIS, T. & SCHERER, C. 2000. Clinical safety of a homeopathic preparation. Biomedical Therapy, 18, 222-225.
- BANNING, M. 2008. Topical diclofenac: clinical effectiveness and current uses in osteoarthritis of the knee and soft tissue injuries. Expert opinion on pharmacotherapy, 9, 2921-9.
- BATTISTI, W. P., WAGER, E., BALTZER, L., BRIDGES, D., CAIRNS, A., CARSWELL, C. I., CITROME, L., GURR, J. A., MOONEY, L. A., MOORE, B.J., PENA, T., SANES-MILLER, C. H., VEITCH, K., WOOLLEY, K. L. & YARKER, Y. E. 2015. Good publication practice for communicating company-sponsored medical research: GPP3. Annals of Internal Medicine, 163, 461-4.
- BIRNESSER, H., OBERBAUM, M., KLEIN, P. & WEISER, M. 2004. The homeopathic preparation Traumeel S compared with NSAIDS for symptomatic treatment of epicondylitis. Journal of Musculoskeletal Research., 8, 119-128.
- BLEAKLEY, C. M., O'CONNOR, S. R., TULLY, M. A., ROCKE, L. G., MACAULEY, D. C., BRADBURY, I., KEEGAN, S. & MCDONOUGH, S. M. 2010. Effect of accelerated rehabilitation on function after ankle sprain: randomised controlled trial. BMJ, 340, c1964.
- BÖHMER, D. & AMBRUS, P. 1992. Treatment of sports injuries with Traumeel ointment: a controlled double-blind study. Biological Therapy, 10, 290-300.
- BRUNNER, E. & MUNZEL, U. 2000. The nonparametric Behrens-Fisher Problem: asymptotic theory and a small-sample approximation. Biometrical Journal, 42, 17-25.
- BRUNNER, U. & MUNZEL, E. 2013. Nichtparametrische Datenanalyse, Berlin, Springer.
- CARCIA, C. R., MARTIN, R. L. & DROUIN, J. M. 2008. Validity of the foot and ankle ability measure in athletes with chronic ankle instability. Journal of Athletic Training, 43, 179-83.
- CHILDS, S. G. 2012. Syndesmotic ankle sprain. Orthopedic Nursing, 31, 177-84.
- COLDITZ, G. A., MILLER, J. N. & MOSTELLER, F. 1988. Measuring gain in the evaluation of medical technology. The probability of a better outcome. International Journal of Technology Assessment in Health Care, 4, 637-42.

- D'AGOSTINO, R. B., CAMPBELL, M. & GREENHOUSE, J. 2006. The Mann—Whitney statistic: continuous use and discovery. Statistics in Medicine, 25, 541-542.
- GONZÁLEZ DE VEGA, C., SPEED, C., WOLFARTH, B. & GONZÁLEZ, J. 2013. Traumeel vs. diclofenac for reducing pain and improving ankle mobility after acute ankle sprain: a multicentre, randomised, blinded, controlled and non-inferiority trial. International Journal of Clinical Practice, 67, 979-989.
- GREEN, T., REFSHAUGE, K., CROSBIE, J. & ADAMS, R. 2001. A randomized controlled trial of a passive accessory joint mobilization on acute ankle inversion sprains. Physical Therapy, 81, 984-94.
- GRIBBLE, P. A., BLEAKLEY, C. M., CAULFIELD, B. M., DOCHERTY, C. L., FOURCHET, F., FONG, D. T., HERTEL, J., HILLER, C. E., KAMINSKI, T. W., MCKEON, P. O., REFSHAUGE, K. M., VERHAGEN, E. A., VICENZINO, B.T., WIKSTROM, E. A. & DELAHUNT, E. 2016. Evidence review for the 2016 International Ankle Consortium consensus statement on the prevalence, impact and long-term consequences of lateral ankle sprains. British Journal of Sports Medicine, 50, 1496-1505.
- HEINE, H. & ANDRÄ, F. 2002. On the anti-inflammatory mechanism of action of an antihomotoxic compound remedy [In German]. Ärztezeitschrift für Naturheilverfahren, 43, 96-104.
- HEUMANN PHARMA GMBH & CO. GENERICA KG, N., GERMANY Diclofenac Heumann Gel. Official summary of product characteristics, 2013.
- HUBBARD, T. J. & CORDOVA, M. 2009. Mechanical instability after an acute lateral ankle sprain. Archives of Physical Medicine and Rehabilitation, 90, 1142-6.
- IVINS, D. 2006. Acute ankle sprain: an update. American Family Physician, 74, 1714-20.
- KIESER, M., FRIEDE, T. & GONDAN, M. 2013. Assessment of statistical significance and clinical relevance. Statistics in Medicine, 32, 1707-19.
- LIN, J., ZHANG, W., JONES, A. & DOHERTY, M. 2004. Efficacy of topical nonsteroidal anti-inflammatory drugs in the treatment of osteoarthritis: meta-analysis of randomised controlled trials. BMJ, 329, 324.
- LUSSIGNOLI, S., BERTANI, S., METELMANN, H., BELLAVITE, P. & CONFORTI, A. 1999. Effect of Traumeel S, a homeopathic formulation, on blood-induced inflammation in rats. Complementary Therapies in Medicine, 7, 225-30.
- MANN, H. B. & WHITNEY, D. R. 1947. On a test of whether one of two random variables is stochastically larger than the other. The Annals of Mathematical Statistics, 18, 50-60.

- MARTIN, R. L., IRRGANG, J. J., BURDETT, R. G., CONTI, S. F. & VAN SWEARINGEN, J. M. 2005. Evidence of validity for the foot and ankle ability measure (FAAM). Foot & Ankle International, 26, 968-83.
- MASON, L., MOORE, R. A., EDWARDS, J. E., DERRY, S. & MCQUAY, H. J. 2004. Topical NSAIDs for acute pain: a meta-analysis. BMC Family Practice, 5, 10.
- MASON, L., MOORE, R. A., EDWARDS, J. E., DERRY, S. & MCQUAY, H. J. 2004. Topical NSAIDs for chronic musculoskeletal pain: systematic review and metaanalysis. BMC Musculoskeletal Disorders, 5, 28.
- MAURER, W., HOTHORN, L. A. & LEHMACHER, W. 1995. Multiple comparisons in drug clinical trials and preclinical assays: a-priori ordered hypotheses. In: VOLLMAR, J. (ed.) Testing Principles in Clinical and Pre-clinical Trials. Stuttgart: G. Fischer.
- MCKAY, G. D., GOLDIE, P. A., PAYNE, W. R. & OAKES, B. W. 2001. Ankle injuries in basketball: injury rate and risk factors. British Journal of Sports Medicine, 35, 103-8.
- MUNZEL, U. & HAUSCHKE, D. 2003. A nonparametric test for proving noninferiority in clinical trials with ordered categorical data. Pharmaceutical Statistics, 2, 31-37.
- O'BRIEN, P. C., ZHANG, D. & BAILEY, K. R. 2005. Semi-parametric and non-parametric methods for clinical trials with incomplete data. Statistics in Medicine, 24, 341-58.
- PREDEL, H. G., KOLL, R., PABST, H., DIETER, R., GALLACCHI, G., GIANNETTI, B., BULITTA, M., HEIDECKER, J. L. & MUELLER, E. A. 2004. Diclofenac patch for topical treatment of acute impact injuries: a randomised, double blind, placebo controlled, multicentre study. British Journal of Sports Medicine, 38, 318-23.
- RAHLFS, V. W., ZIMMERMANN, H. & LEES, K. R. 2014. Effect size measures and their relationships in stroke studies. Stroke, 45, 627-33.
- ROTHMANN, M. D., MILLER, J. N., WIENS, B. L. & CHAN, I. S. 2011. Design and Analysis of Non-Inferiority Trials, Boca Raton, FL, Chapman & Hall.
- SCHNEIDER, C. 2011. Traumeel: an emerging option to nonsteroidal antiinflammatory drugs in the management of acute musculoskeletal injuries. International Journal of General Medicine, 4, 225-234.
- SCHNEIDER, C., KLEIN, P., STOLT, P. & OBERBAUM, M. 2005. A homeopathic ointment preparation compared with 1% diclofenac gel for acute symptomatic treatment of tendinopathy. Explore (NY), 1, 446-52.

41 of 75

- SCHNEIDER, C., SCHNEIDER, B., HANISCH, J. & VAN HASELEN, R. 2008. The role of a homoeopathic preparation compared with conventional therapy in the treatment of injuries: an observational cohort study. Complementary Therapies in Medicine, 16, 22-27.
- SCHOMACHER, J. 2008. Gütekriterien der visuellen Analogskala zur Schmerzbewertung: quality criteria of the visual analogue scale for pain assessment. Physioscience, 4, 125-133.
- SIMON, L. S., GRIERSON, L. M., NASEER, Z., BOOKMAN, A. A. & ZEV SHAINHOUSE, J. 2009. Efficacy and safety of topical diclofenac containing dimethyl sulfoxide (DMSO) compared with those of topical placebo, DMSO vehicle and oral diclofenac for knee osteoarthritis. Pain, 143, 238-45.
- SPRENT, P. & SMEETON, N. C. 2001. Applied Nonparametric Statistical Methods, Boca Raton, Chapman and Hall.
- TAYLOR, R. S., FOTOPOULOS, G. & MAIBACH, H. 2011. Safety profile of topical diclofenac: a meta-analysis of blinded, randomized, controlled trials in musculoskeletal conditions. Current Medical Research and Opinion, 27, 605-22.
- THIEL, W. & BORHO, B. 1994. The treatment of recent traumatic blood effusions of the knee joint. Biological Therapy, 12, 242-248.
- TIEMSTRA, J. D. 2012. Update on acute ankle sprains. American Family Physician, 85, 1170-6.
- TUBACH, F., RAVAUD, P., BARON, G., FALISSARD, B., LOGEART, I., BELLAMY, N., BOMBARDIER, C., FELSON, D., HOCHBERG, M., VAN DER HEIJDE, D. & DOUGADOS, M. 2005. Evaluation of clinically relevant changes in patient reported outcomes in knee and hip osteoarthritis: the minimal clinically important improvement. Annals of the Rheumatic Diseases, 64, 29-33.
- TUBACH, F., RAVAUD, P., BARON, G., FALISSARD, B., LOGEART, I., BELLAMY, N., BOMBARDIER, C., FELSON, D., HOCHBERG, M., VAN DER HEIJDE, D. & DOUGADOS, M. 2005. Evaluation of clinically relevant states in patient reported outcomes in knee and hip osteoarthritis: the patient acceptable symptom state. Annals of the Rheumatic Diseases, 64, 34-7.
- WEXLER, R. K. 1998. The injured ankle. American Family Physician, 57, 474-80.
- WILCOXON, F. 1945. Individual comparisons by ranking methods. Biometrics Bulletin, 1, 80-83.
- WOLFE, M. W., UHL, T. L., MATTACOLA, C. G. & MCCLUSKEY, L. C. 2001. Management of ankle sprains. American Family Physician, 63, 93-104.

- ZACHER, J., ALTMAN, R., BELLAMY, N., BRUHLMANN, P., DA SILVA, J., HUSKISSON, E. & TAYLOR, R. S. 2008. Topical diclofenac and its role in pain and inflammation: an evidence-based review. Current Medical Research and Opinion, 24, 925-50.
- ZELL, J., CONNERT, W. D., MAU, J. & FEUERSTAKE, G. 1988. Behandlung von Sprunggelenksdistorsionen: Doppelblindstudie zum Wirksamkeitsnachweis eines homöopathischen Salbenpräparats. Fortschritte der Medizin, 106, 96-100.

#### 13. APPENDIX

### 13.1 BDRM Decisions

#### 13.1.1 Problem Cases

Besides the 'issue' cases addressed in C1502 Study Protocol Version 4.0 (3 February 2020) and in the Amendment Summary Document for Substantial protocol Changes (3 February 2020), no other problem cases were identified. For details see section 8 *Changes to the Protocol*.

### 13.1.2 Other Decisions

Day 7 was introduced as additional endpoint in the chain of *a priori* ordered hypotheses (hypotheses no. 3 and no. 4). This addition was implemented as per BDRM decision in order to avoid lack of assay sensitivity at the very early stage of the ankle joint injury (C1502\_MTG\_NOTES\_BDRM\_09MAR2021\_20210324).

### 13.2 Individual Dataset Assignment

The following table shows the individual dataset assignment based on the hardlock transfer for 'non-issue' patients (in Table 1) and 'issue' patients (in Table 2) (see section 8 *Changes to the Protocol*).

Table 1: Dataset Assignment, Status: Hardlock Transfer, 'Non-issue' Patients (n = 625)

| PATID | RANDOM<br>NUMBER | SAFETY | FAS | PP |
|----------|------------------|--------|-----|----|
| 4902-001 | 1073 | 1 | 1 | 1 |
| 4902-002 | 1074 | 1 | 1 | 1 |
| 4902-003 | 1075 | 1 | 1 | 1 |
| 4902-004 | 1076 | 1 | 1 | 1 |
| 4902-005 | 1077 | 1 | 1 | 1 |
| 4902-006 | 1078 | 1 | 1 | 1 |
| 4902-007 | 1079 | 1 | 1 | 0 |
| 4902-008 | 1080 | 1 | 1 | 1 |
| 4902-009 | 1217 | 1 | 1 | 1 |
| 4902-010 | 1218 | 1 | 1 | 1 |
| 4902-011 | 1219 | 1 | 1 | 1 |
| 4902-012 | 1220 | 1 | 1 | 1 |
| 4902-013 | 1221 | 1 | 1 | 1 |
| 4902-014 | 1222 | 1 | 1 | 1 |
| 4902-015 | 1223 | 1 | 1 | 1 |
| 4902-016 | 1224 | 1 | 1 | 1 |
| 4902-017 | 1561 | 1 | 1 | 0 |
| 4902-018 | 1562 | 1 | 1 | 1 |
| 4902-019 | 1563 | 1 | 1 | 1 |

| PATID | RANDOM<br>NUMBER | SAFETY | FAS | PP |
|----------|------------------|--------|-----|----|
| 4902-020 | 1564 | 1 | 1 | 1 |
| 4902-021 | 1565 | 1 | 1 | 1 |
| 4902-022 | 1568 | 1 | 1 | 1 |
| 4902-023 | 1566 | 1 | 1 | 1 |
| 4902-024 | 1567 | 1 | 1 | 1 |
| 4902-025 | 1729 | 1 | 1 | 1 |
| 4902-026 | 1730 | 1 | 1 | 1 |
| 4903-001 | 1089 | 1 | 1 | 0 |
| 4903-002 | 1090 | 1 | 1 | 1 |
| 4903-003 | 1091 | 1 | 1 | 1 |
| 4903-004 | 1092 | 1 | 1 | 1 |
| 4903-005 | 1093 | 1 | 1 | 1 |
| 4903-006 | 1094 | 1 | 1 | 1 |
| 4905-009 | 1457 | 1 | 0 | 0 |
| 4905-010 | 1458 | 1 | 1 | 1 |
| 4906-001 | 1049 | 1 | 1 | 1 |
| 4906-002 | 1050 | 1 | 1 | 1 |
| 4906-003 | 1051 | 1 | 1 | 1 |
| 4906-004 | 1052 | 1 | 1 | 1 |
| 4906-005 | 1053 | 1 | 1 | 1 |
| 4906-006 | 1054 | 1 | 1 | 1 |
| 4906-007 | 1055 | 1 | 1 | 1 |
| 4906-008 | 1056 | 1 | 1 | 1 |
| 4906-009 | 1233 | 1 | 1 | 1 |
| 4906-010 | 1234 | 1 | 1 | 1 |
| 4906-011 | 1235 | 1 | 1 | 1 |
| 4906-012 | 1236 | 1 | 1 | 1 |
| 4906-013 | 1237 | 1 | 1 | 1 |
| 4906-014 | 1238 | 1 | 1 | 1 |
| 4906-015 | 1239 | 1 | 1 | 1 |
| 4906-016 | 1240 | 1 | 1 | 1 |
| 4906-017 | 1385 | 1 | 1 | 1 |
| 4906-018 | 1386 | 1 | 1 | 1 |
| 4906-019 | 1387 | 1 | 1 | 1 |
| 4906-020 | 1388 | 1 | 1 | 1 |
| 4906-021 | 1389 | 1 | 1 | 1 |
| 4906-022 | 1390 | 1 | 1 | 1 |
| 4906-023 | 1391 | 1 | 1 | 1 |
| 4906-024 | 1392 | 1 | 1 | 1 |
| 4906-025 | 1441 | 1 | 1 | 1 |
| 4906-026 | 1442 | 1 | 1 | 1 |
| 4906-027 | 1443 | 1 | 1 | 1 |

| PATID | RANDOM<br>NUMBER | SAFETY | FAS | PP |
|----------|------------------|--------|-----|----|
| 4906-028 | 1444 | 1 | 1 | 1 |
| 4906-029 | 1445 | 1 | 1 | 1 |
| 4906-030 | 1446 | 1 | 1 | 1 |
| 4906-031 | 1447 | 1 | 1 | 1 |
| 4906-032 | 1448 | 1 | 1 | 1 |
| 4906-033 | 1577 | 1 | 1 | 1 |
| 4906-034 | 1578 | 1 | 1 | 1 |
| 4906-035 | 1579 | 1 | 1 | 1 |
| 4906-036 | 1580 | 1 | 1 | 1 |
| 4906-037 | 1581 | 1 | 1 | 1 |
| 4906-038 | 1582 | 1 | 1 | 1 |
| 4906-039 | 1583 | 1 | 1 | 1 |
| 4906-040 | 1584 | 1 | 1 | 1 |
| 4906-041 | 1649 | 1 | 1 | 1 |
| 4906-042 | 1650 | 1 | 1 | 1 |
| 4906-043 | 1651 | 1 | 1 | 1 |
| 4906-044 | 3009 | 1 | 1 | 1 |
| 4906-045 | 3010 | 1 | 1 | 1 |
| 4906-046 | 3011 | 1 | 1 | 1 |
| 4906-047 | 3012 | 1 | 1 | 1 |
| 4906-048 | 3109 | 1 | 1 | 1 |
| 4906-049 | 3110 | 1 | 1 | 1 |
| 4906-050 | 3111 | 1 | 1 | 1 |
| 4906-051 | 3112 | 1 | 1 | 1 |
| 4906-052 | 3149 | 1 | 1 | 1 |
| 4907-001 | 1009 | 1 | 1 | 1 |
| 4907-002 | 1010 | 1 | 1 | 1 |
| 4907-003 | 1011 | 1 | 1 | 1 |
| 4907-004 | 1012 | 1 | 1 | 1 |
| 4907-005 | 1013 | 1 | 1 | 1 |
| 4907-006 | 1014 | 1 | 1 | 1 |
| 4907-007 | 1015 | 1 | 1 | 1 |
| 4907-008 | 1016 | 1 | 1 | 1 |
| 4907-009 | 1161 | 1 | 1 | 1 |
| 4907-010 | 1162 | 1 | 1 | 1 |
| 4907-011 | 1163 | 1 | 1 | 1 |
| 4907-012 | 1164 | 1 | 1 | 1 |
| 4907-013 | 1165 | 1 | 1 | 1 |
| 4907-014 | 1166 | 1 | 1 | 1 |
| 4907-015 | 1167 | 1 | 1 | 1 |
| 4907-016 | 1168 | 1 | 1 | 1 |
| 4907-017 | 1329 | 1 | 1 | 1 |

| PATID | RANDOM<br>NUMBER | SAFETY | FAS | PP |
|----------|------------------|--------|-----|----|
| 4907-018 | 1330 | 1 | 1 | 1 |
| 4907-019 | 1331 | 1 | 1 | 1 |
| 4907-020 | 1332 | 1 | 1 | 1 |
| 4907-021 | 1333 | 1 | 1 | 1 |
| 4907-022 | 1334 | 1 | 1 | 1 |
| 4907-023 | 1335 | 1 | 1 | 1 |
| 4907-024 | 1336 | 1 | 1 | 1 |
| 4907-025 | 1489 | 1 | 1 | 1 |
| 4907-026 | 1490 | 1 | 1 | 1 |
| 4907-027 | 1491 | 1 | 1 | 1 |
| 4907-028 | 1492 | 1 | 1 | 1 |
| 4907-029 | 1493 | 1 | 1 | 1 |
| 4907-030 | 1494 | 1 | 1 | 1 |
| 4907-031 | 1495 | 1 | 1 | 1 |
| 4907-032 | 1496 | 1 | 1 | 1 |
| 4907-033 | 1537 | 1 | 1 | 1 |
| 4907-034 | 1538 | 1 | 1 | 1 |
| 4907-035 | 1539 | 1 | 1 | 1 |
| 4907-036 | 1540 | 1 | 1 | 1 |
| 4907-037 | 1541 | 1 | 1 | 1 |
| 4907-038 | 1542 | 1 | 1 | 1 |
| 4907-039 | 1543 | 1 | 1 | 1 |
| 4907-040 | 1544 | 1 | 1 | 1 |
| 4907-041 | 1673 | 1 | 1 | 1 |
| 4907-042 | 1674 | 1 | 1 | 1 |
| 4907-043 | 1675 | 1 | 0 | 0 |
| 4907-044 | 1676 | 1 | 1 | 1 |
| 4907-045 | 1677 | 1 | 1 | 1 |
| 4907-046 | 1678 | 1 | 1 | 1 |
| 4907-047 | 1679 | 1 | 1 | 1 |
| 4907-048 | 3105 | 1 | 1 | 1 |
| 4907-049 | 3106 | 1 | 1 | 1 |
| 4907-050 | 3107 | 1 | 1 | 1 |
| 4907-051 | 3108 | 1 | 1 | 1 |
| 4907-052 | 3309 | 1 | 1 | 1 |
| 4908-001 | 1145 | 1 | 1 | 1 |
| 4908-002 | 1146 | 1 | 1 | 1 |
| 4908-003 | 1147 | 1 | 1 | 1 |
| 4908-004 | 1148 | 1 | 1 | 1 |
| 4908-005 | 1149 | 1 | 1 | 1 |
| 4908-006 | 1151 | 1 | 1 | 1 |
| 4908-007 | 1150 | 1 | 1 | 1 |

| PATID | RANDOM<br>NUMBER | SAFETY | FAS | PP |
|----------|------------------|--------|-----|----|
| 4908-008 | 1152 | 1 | 1 | 1 |
| 4908-009 | 1345 | 1 | 1 | 1 |
| 4908-010 | 1346 | 1 | 1 | 1 |
| 4908-011 | 1347 | 1 | 1 | 1 |
| 4908-012 | 1348 | 1 | 1 | 1 |
| 4908-013 | 1349 | 1 | 1 | 1 |
| 4908-014 | 1350 | 1 | 1 | 1 |
| 4908-015 | 1351 | 1 | 1 | 1 |
| 4908-016 | 1352 | 1 | 1 | 1 |
| 4908-017 | 1585 | 1 | 1 | 1 |
| 4908-018 | 1586 | 1 | 1 | 1 |
| 4908-019 | 1587 | 1 | 1 | 1 |
| 4908-020 | 1588 | 1 | 1 | 1 |
| 4908-021 | 1589 | 1 | 1 | 1 |
| 4908-022 | 1590 | 1 | 1 | 1 |
| 4908-023 | 1591 | 1 | 1 | 1 |
| 4908-024 | 1592 | 1 | 1 | 1 |
| 4908-025 | 1633 | 1 | 1 | 1 |
| 4908-026 | 1634 | 1 | 1 | 1 |
| 4908-027 | 1635 | 1 | 1 | 1 |
| 4908-028 | 1636 | 1 | 1 | 1 |
| 4908-029 | 1637 | 1 | 1 | 1 |
| 4908-030 | 1638 | 1 | 1 | 1 |
| 4908-031 | 1639 | 1 | 1 | 1 |
| 4908-032 | 1640 | 1 | 1 | 1 |
| 4908-033 | 3073 | 1 | 1 | 1 |
| 4909-001 | 1041 | 1 | 1 | 1 |
| 4909-002 | 1042 | 1 | 1 | 1 |
| 4909-011 | 1155 | 1 | 1 | 1 |
| 4909-012 | 1156 | 1 | 1 | 1 |
| 4909-015 | 1159 | 1 | 1 | 1 |
| 4909-016 | 1160 | 1 | 1 | 1 |
| 4909-017 | 1417 | 1 | 1 | 1 |
| 4909-018 | 1418 | 1 | 1 | 1 |
| 4909-019 | 1419 | 1 | 1 | 1 |
| 4909-036 | 1660 | 1 | 1 | 1 |
| 4909-037 | 1661 | 1 | 1 | 1 |
| 4909-038 | 1662 | 1 | 1 | 1 |
| 4909-039 | 1663 | 1 | 1 | 1 |
| 4909-040 | 1664 | 1 | 1 | 1 |
| 4909-041 | 3013 | 1 | 1 | 1 |
| 4909-042 | 3014 | 1 | 1 | 1 |

| PATID | RANDOM<br>NUMBER | SAFETY | FAS | PP |
|----------|------------------|--------|-----|----|
| 4909-043 | 3015 | 1 | 1 | 1 |
| 4909-044 | 3016 | 1 | 1 | 1 |
| 4909-045 | 3133 | 1 | 1 | 1 |
| 4909-046 | 3134 | 1 | 1 | 1 |
| 4909-047 | 3135 | 1 | 1 | 1 |
| 4910-046 | 1646 | 1 | 1 | 1 |
| 4910-047 | 1647 | 1 | 1 | 1 |
| 4910-048 | 1648 | 1 | 1 | 1 |
| 4910-049 | 1737 | 1 | 1 | 1 |
| 4910-050 | 1738 | 1 | 1 | 1 |
| 4910-051 | 1739 | 1 | 1 | 1 |
| 4910-052 | 1740 | 1 | 1 | 1 |
| 4910-053 | 1741 | 1 | 1 | 1 |
| 4910-054 | 1742 | 1 | 1 | 1 |
| 4910-055 | 1743 | 1 | 1 | 1 |
| 4910-056 | 1744 | 1 | 1 | 1 |
| 4910-057 | 3077 | 1 | 1 | 1 |
| 4910-058 | 3078 | 1 | 1 | 1 |
| 4910-059 | 3079 | 1 | 1 | 1 |
| 4910-060 | 3080 | 1 | 1 | 1 |
| 4910-061 | 3153 | 1 | 1 | 1 |
| 4910-062 | 3154 | 1 | 1 | 1 |
| 4910-063 | 3155 | 1 | 1 | 1 |
| 4910-064 | 3156 | 1 | 1 | 1 |
| 4910-065 | 3189 | 1 | 1 | 1 |
| 4910-066 | 3190 | 1 | 1 | 1 |
| 4910-067 | 3191 | 1 | 1 | 1 |
| 4910-068 | 3192 | 1 | 1 | 1 |
| 4910-069 | 3193 | 1 | 1 | 1 |
| 4910-070 | 3194 | 1 | 1 | 1 |
| 4910-071 | 3195 | 1 | 1 | 1 |
| 4910-072 | 3196 | 1 | 1 | 1 |
| 4910-073 | 3209 | 1 | 1 | 1 |
| 4910-074 | 3210 | 1 | 1 | 1 |
| 4910-075 | 3211 | 1 | 1 | 1 |
| 4910-076 | 3212 | 1 | 1 | 1 |
| 4910-077 | 3261 | 1 | 1 | 1 |
| 4910-078 | 3262 | 1 | 1 | 1 |
| 4910-079 | 3263 | 1 | 1 | 1 |
| 4910-080 | 3264 | 1 | 1 | 1 |
| 4910-081 | 3265 | 1 | 1 | 1 |
| 4910-082 | 3266 | 1 | 1 | 1 |

| PATID | RANDOM<br>NUMBER | SAFETY | FAS | PP |
|----------|------------------|--------|-----|----|
| 4910-083 | 3267 | 1 | 1 | 1 |
| 4910-084 | 3268 | 1 | 1 | 1 |
| 4910-085 | 3293 | 1 | 1 | 1 |
| 4910-086 | 3294 | 1 | 1 | 1 |
| 4910-087 | 3295 | 1 | 1 | 1 |
| 4910-088 | 3296 | 1 | 1 | 1 |
| 4910-089 | 3297 | 1 | 1 | 1 |
| 4910-090 | 3298 | 1 | 1 | 1 |
| 4911-006 | 3053 | 1 | 1 | 1 |
| 4911-007 | 3054 | 1 | 1 | 0 |
| 4911-008 | 3055 | 1 | 1 | 1 |
| 4911-009 | 3056 | 1 | 1 | 1 |
| 4911-010 | 3085 | 1 | 1 | 1 |
| 4911-011 | 3086 | 1 | 1 | 1 |
| 4911-012 | 3087 | 1 | 1 | 1 |
| 4912-001 | 1017 | 1 | 1 | 1 |
| 4912-002 | 1018 | 1 | 1 | 1 |
| 4912-003 | 1019 | 1 | 1 | 1 |
| 4915-001 | 1025 | 1 | 1 | 1 |
| 4915-002 | 1026 | 1 | 1 | 1 |
| 4915-003 | 1027 | 1 | 1 | 1 |
| 4915-004 | 1028 | 1 | 1 | 1 |
| 4915-005 | 1029 | 1 | 1 | 1 |
| 4915-006 | 1030 | 1 | 1 | 1 |
| 4915-007 | 1031 | 1 | 1 | 1 |
| 4915-008 | 1032 | 1 | 1 | 1 |
| 4915-009 | 1169 | 1 | 1 | 1 |
| 4915-010 | 1170 | 1 | 1 | 1 |
| 4915-011 | 1171 | 1 | 1 | 1 |
| 4915-012 | 1172 | 1 | 1 | 1 |
| 4915-013 | 1173 | 1 | 1 | 1 |
| 4915-014 | 1174 | 1 | 1 | 1 |
| 4915-015 | 1175 | 1 | 1 | 1 |
| 4915-016 | 1176 | 1 | 1 | 1 |
| 4915-017 | 1193 | 1 | 1 | 1 |
| 4915-018 | 1194 | 1 | 1 | 1 |
| 4915-019 | 1195 | 1 | 1 | 1 |
| 4915-020 | 1196 | 1 | 1 | 1 |
| 4915-021 | 1197 | 1 | 1 | 1 |
| 4915-022 | 1198 | 1 | 1 | 1 |
| 4915-023 | 1199 | 1 | 1 | 1 |
| 4915-024 | 1200 | 1 | 1 | 1 |

| PATID | RANDOM<br>NUMBER | SAFETY | FAS | PP |
|----------|------------------|--------|-----|----|
| 4915-025 | 1201 | 1 | 1 | 1 |
| 4915-026 | 1202 | 1 | 1 | 1 |
| 4915-027 | 1203 | 1 | 1 | 1 |
| 4915-028 | 1204 | 1 | 1 | 1 |
| 4915-029 | 1205 | 1 | 1 | 1 |
| 4915-030 | 1206 | 1 | 1 | 1 |
| 4915-031 | 1207 | 1 | 1 | 1 |
| 4915-032 | 1208 | 1 | 1 | 1 |
| 4915-033 | 1225 | 1 | 1 | 1 |
| 4915-034 | 1226 | 1 | 1 | 1 |
| 4915-035 | 1227 | 1 | 1 | 1 |
| 4915-036 | 1228 | 1 | 1 | 1 |
| 4915-037 | 1229 | 1 | 1 | 1 |
| 4915-038 | 1230 | 1 | 1 | 1 |
| 4915-039 | 1231 | 1 | 1 | 1 |
| 4915-040 | 1232 | 1 | 1 | 1 |
| 4915-041 | 1305 | 1 | 1 | 1 |
| 4915-042 | 1306 | 1 | 1 | 1 |
| 4915-043 | 1307 | 1 | 1 | 1 |
| 4915-044 | 1308 | 1 | 1 | 1 |
| 4915-045 | 1309 | 1 | 1 | 1 |
| 4915-046 | 1310 | 1 | 1 | 1 |
| 4915-047 | 1311 | 1 | 1 | 1 |
| 4915-048 | 1312 | 1 | 1 | 1 |
| 4915-049 | 1401 | 1 | 1 | 1 |
| 4915-050 | 1402 | 1 | 1 | 1 |
| 4915-051 | 1403 | 1 | 1 | 1 |
| 4915-052 | 1404 | 1 | 1 | 1 |
| 4915-053 | 1405 | 1 | 1 | 1 |
| 4915-054 | 1406 | 1 | 1 | 1 |
| 4915-055 | 1407 | 1 | 1 | 1 |
| 4915-056 | 1408 | 1 | 1 | 1 |
| 4915-057 | 3121 | 1 | 1 | 1 |
| 4915-058 | 3122 | 1 | 1 | 1 |
| 4915-059 | 3123 | 1 | 1 | 1 |
| 4915-060 | 3124 | 1 | 1 | 1 |
| 4915-061 | 3126 | 1 | 1 | 1 |
| 4915-062 | 3125 | 1 | 1 | 1 |
| 4915-063 | 3127 | 1 | 1 | 1 |
| 4915-064 | 3128 | 1 | 1 | 1 |
| 4915-065 | 3129 | 1 | 1 | 1 |
| 4915-066 | 3130 | 1 | 1 | 1 |

| PATID | RANDOM<br>NUMBER | SAFETY | FAS | PP |
|----------|------------------|--------|-----|----|
| 4915-067 | 3131 | 1 | 1 | 1 |
| 4915-068 | 3132 | 1 | 1 | 1 |
| 4915-069 | 3177 | 1 | 1 | 1 |
| 4915-070 | 3178 | 1 | 1 | 1 |
| 4915-071 | 3179 | 1 | 1 | 1 |
| 4915-072 | 3180 | 1 | 1 | 1 |
| 4915-073 | 3181 | 1 | 1 | 1 |
| 4915-074 | 3182 | 1 | 1 | 1 |
| 4915-075 | 3183 | 1 | 1 | 1 |
| 4915-076 | 3184 | 1 | 1 | 1 |
| 4915-077 | 3185 | 1 | 1 | 1 |
| 4915-078 | 3186 | 1 | 1 | 1 |
| 4915-079 | 3187 | 1 | 1 | 1 |
| 4915-080 | 3188 | 1 | 1 | 1 |
| 4915-081 | 3245 | 1 | 1 | 1 |
| 4915-082 | 3246 | 1 | 1 | 1 |
| 4915-083 | 3247 | 1 | 1 | 1 |
| 4915-084 | 3248 | 1 | 1 | 1 |
| 4915-085 | 3249 | 1 | 1 | 1 |
| 4915-086 | 3250 | 1 | 1 | 1 |
| 4915-087 | 3251 | 1 | 1 | 1 |
| 4915-088 | 3252 | 1 | 1 | 1 |
| 4915-089 | 3253 | 1 | 1 | 1 |
| 4915-090 | 3254 | 1 | 1 | 1 |
| 4915-091 | 3255 | 1 | 1 | 1 |
| 4915-092 | 3256 | 1 | 1 | 1 |
| 4915-093 | 3317 | 1 | 1 | 1 |
| 4915-094 | 3318 | 1 | 1 | 1 |
| 4915-095 | 3319 | 1 | 1 | 1 |
| 4915-096 | 3320 | 1 | 1 | 1 |
| 4915-097 | 3321 | 1 | 1 | 1 |
| 4915-098 | 3322 | 1 | 1 | 1 |
| 4915-099 | 3323 | 1 | 1 | 1 |
| 4915-100 | 3324 | 1 | 1 | 1 |
| 4918-015 | 1319 | 1 | 1 | 1 |
| 4918-016 | 1320 | 1 | 1 | 1 |
| 4918-017 | 1513 | 1 | 1 | 1 |
| 4918-019 | 1515 | 1 | 1 | 1 |
| 4918-020 | 1516 | 1 | 1 | 1 |
| 4918-021 | 1517 | 1 | 1 | 1 |
| 4918-022 | 1518 | 1 | 1 | 1 |
| 4918-023 | 1519 | 1 | 1 | 1 |

| PATID | RANDOM<br>NUMBER | SAFETY | FAS | PP |
|----------|------------------|--------|-----|----|
| 4918-024 | 1520 | 1 | 1 | 1 |
| 4918-025 | 1601 | 1 | 1 | 1 |
| 4918-026 | 1602 | 1 | 1 | 1 |
| 4918-027 | 1603 | 1 | 1 | 1 |
| 4918-028 | 1604 | 1 | 1 | 1 |
| 4918-029 | 1605 | 1 | 1 | 1 |
| 4918-030 | 1606 | 1 | 1 | 1 |
| 4918-031 | 1607 | 1 | 1 | 1 |
| 4918-032 | 3017 | 1 | 1 | 1 |
| 4918-033 | 3018 | 1 | 1 | 1 |
| 4918-034 | 3019 | 1 | 1 | 1 |
| 4918-035 | 3020 | 1 | 1 | 1 |
| 4918-036 | 3113 | 1 | 1 | 1 |
| 4919-001 | 1033 | 1 | 1 | 1 |
| 4919-002 | 1034 | 1 | 1 | 1 |
| 4919-003 | 1035 | 1 | 1 | 1 |
| 4919-004 | 1036 | 1 | 1 | 1 |
| 4919-005 | 1037 | 1 | 1 | 1 |
| 4919-006 | 1038 | 1 | 1 | 1 |
| 4919-007 | 1039 | 1 | 1 | 1 |
| 4919-008 | 1040 | 1 | 1 | 1 |
| 4919-009 | 1185 | 1 | 1 | 1 |
| 4919-010 | 1186 | 1 | 1 | 1 |
| 4919-011 | 1187 | 1 | 1 | 1 |
| 4919-012 | 1188 | 1 | 1 | 1 |
| 4919-013 | 1189 | 1 | 1 | 1 |
| 4919-014 | 1190 | 1 | 1 | 1 |
| 4919-015 | 1191 | 1 | 1 | 1 |
| 4919-016 | 1192 | 1 | 1 | 1 |
| 4919-017 | 1209 | 1 | 1 | 1 |
| 4919-018 | 1210 | 1 | 1 | 1 |
| 4919-019 | 1211 | 1 | 1 | 1 |
| 4919-020 | 1212 | 1 | 1 | 1 |
| 4919-021 | 1213 | 1 | 1 | 1 |
| 4919-022 | 1214 | 1 | 1 | 1 |
| 4919-023 | 1215 | 1 | 1 | 1 |
| 4919-024 | 1216 | 1 | 1 | 1 |
| 4919-025 | 1257 | 1 | 1 | 1 |
| 4919-026 | 1258 | 1 | 1 | 1 |
| 4919-027 | 1259 | 1 | 1 | 1 |
| 4919-028 | 1260 | 1 | 1 | 1 |
| 4919-029 | 1261 | 1 | 1 | 1 |

| PATID | RANDOM<br>NUMBER | SAFETY | FAS | PP |
|----------|------------------|--------|-----|----|
| 4919-030 | 1262 | 1 | 1 | 1 |
| 4919-031 | 1263 | 1 | 1 | 1 |
| 4919-032 | 1264 | 1 | 1 | 1 |
| 4919-033 | 1281 | 1 | 1 | 1 |
| 4919-034 | 1282 | 1 | 1 | 1 |
| 4919-035 | 1283 | 1 | 1 | 1 |
| 4919-036 | 1284 | 1 | 1 | 1 |
| 4919-037 | 1285 | 1 | 1 | 1 |
| 4919-038 | 1286 | 1 | 1 | 1 |
| 4919-039 | 1287 | 1 | 1 | 1 |
| 4919-040 | 1288 | 1 | 1 | 1 |
| 4919-041 | 1409 | 1 | 1 | 1 |
| 4919-042 | 1410 | 1 | 1 | 1 |
| 4919-043 | 1411 | 1 | 1 | 1 |
| 4919-044 | 1412 | 1 | 1 | 1 |
| 4919-045 | 1413 | 1 | 1 | 1 |
| 4919-046 | 1414 | 1 | 1 | 1 |
| 4919-047 | 1415 | 1 | 1 | 1 |
| 4919-048 | 1416 | 1 | 1 | 1 |
| 4919-049 | 1481 | 1 | 1 | 1 |
| 4919-050 | 1482 | 1 | 1 | 1 |
| 4919-051 | 1483 | 1 | 1 | 1 |
| 4919-052 | 1484 | 1 | 1 | 1 |
| 4919-053 | 1485 | 1 | 1 | 1 |
| 4919-054 | 1486 | 1 | 1 | 1 |
| 4919-055 | 1487 | 1 | 1 | 1 |
| 4919-056 | 1488 | 1 | 1 | 1 |
| 4919-057 | 3093 | 1 | 1 | 1 |
| 4919-058 | 3094 | 1 | 1 | 1 |
| 4919-059 | 3095 | 1 | 1 | 1 |
| 4919-060 | 3096 | 1 | 1 | 1 |
| 4919-061 | 3097 | 1 | 1 | 1 |
| 4919-062 | 3098 | 1 | 1 | 1 |
| 4919-063 | 3099 | 1 | 1 | 1 |
| 4919-064 | 3100 | 1 | 1 | 1 |
| 4919-065 | 3101 | 1 | 1 | 1 |
| 4919-066 | 3102 | 1 | 1 | 1 |
| 4919-067 | 3103 | 1 | 1 | 1 |
| 4919-068 | 3104 | 1 | 1 | 1 |
| 4919-069 | 3161 | 1 | 1 | 1 |
| 4919-070 | 3162 | 1 | 1 | 1 |
| 4919-071 | 3163 | 1 | 1 | 1 |

| PATID | RANDOM<br>NUMBER | SAFETY | FAS | PP |
|----------|------------------|--------|-----|----|
| 4919-072 | 3164 | 1 | 1 | 1 |
| 4919-073 | 3165 | 1 | 1 | 1 |
| 4919-074 | 3166 | 1 | 1 | 1 |
| 4919-075 | 3167 | 1 | 1 | 1 |
| 4919-076 | 3168 | 1 | 1 | 1 |
| 4919-077 | 3169 | 1 | 1 | 1 |
| 4919-078 | 3170 | 1 | 1 | 1 |
| 4919-079 | 3171 | 1 | 1 | 1 |
| 4919-080 | 3172 | 1 | 1 | 1 |
| 4919-081 | 3233 | 1 | 1 | 1 |
| 4919-082 | 3234 | 1 | 1 | 1 |
| 4919-083 | 3235 | 1 | 1 | 1 |
| 4919-084 | 3236 | 1 | 1 | 1 |
| 4919-085 | 3237 | 1 | 1 | 1 |
| 4919-086 | 3238 | 1 | 1 | 1 |
| 4920-001 | 1121 | 1 | 1 | 1 |
| 4920-002 | 1122 | 1 | 1 | 1 |
| 4920-003 | 1123 | 1 | 1 | 1 |
| 4920-004 | 1124 | 1 | 1 | 1 |
| 4920-005 | 1125 | 1 | 1 | 1 |
| 4920-006 | 1126 | 1 | 1 | 1 |
| 4920-007 | 1127 | 1 | 1 | 1 |
| 4920-008 | 1128 | 1 | 1 | 1 |
| 4920-009 | 1297 | 1 | 1 | 1 |
| 4920-010 | 1298 | 1 | 1 | 1 |
| 4920-011 | 1299 | 1 | 1 | 1 |
| 4920-012 | 1300 | 1 | 1 | 1 |
| 4920-013 | 1301 | 1 | 1 | 1 |
| 4920-014 | 1302 | 1 | 1 | 1 |
| 4920-015 | 1303 | 1 | 1 | 1 |
| 4921-002 | 1106 | 1 | 1 | 1 |
| 4921-011 | 1291 | 1 | 1 | 1 |
| 4921-012 | 1292 | 1 | 1 | 1 |
| 4921-013 | 1293 | 1 | 1 | 1 |
| 4921-016 | 1296 | 1 | 1 | 1 |
| 4921-020 | 1373 | 1 | 1 | 1 |
| 4921-021 | 1374 | 1 | 1 | 1 |
| 4921-022 | 1369 | 1 | 1 | 1 |
| 4921-023 | 1375 | 1 | 1 | 1 |
| 4921-024 | 1376 | 1 | 1 | 1 |
| 4921-025 | 1465 | 1 | 1 | 1 |
| 4921-027 | 1467 | 1 | 1 | 1 |

| PATID | RANDOM<br>NUMBER | SAFETY | FAS | PP |
|----------|------------------|--------|-----|----|
| 4921-029 | 1469 | 1 | 1 | 1 |
| 4921-039 | 1575 | 1 | 1 | 1 |
| 4921-048 | 1624 | 1 | 1 | 1 |
| 4921-049 | 1689 | 1 | 1 | 1 |
| 4921-050 | 1690 | 1 | 1 | 1 |
| 4921-055 | 1695 | 1 | 1 | 1 |
| 4921-056 | 1696 | 1 | 1 | 1 |
| 4921-057 | 3021 | 1 | 1 | 1 |
| 4921-058 | 3022 | 1 | 1 | 1 |
| 4921-059 | 3023 | 1 | 1 | 1 |
| 4921-060 | 3024 | 1 | 1 | 1 |
| 4921-061 | 3145 | 1 | 1 | 1 |
| 4921-062 | 3146 | 1 | 1 | 1 |
| 4921-063 | 3147 | 1 | 1 | 1 |
| 4921-064 | 3148 | 1 | 1 | 1 |
| 4923-030 | 1630 | 1 | 1 | 1 |
| 4923-031 | 1631 | 1 | 1 | 1 |
| 4923-032 | 1632 | 1 | 1 | 1 |
| 4923-033 | 1721 | 1 | 1 | 1 |
| 4923-034 | 1722 | 1 | 1 | 1 |
| 4923-035 | 1723 | 1 | 1 | 1 |
| 4923-036 | 1724 | 1 | 1 | 1 |
| 4923-037 | 1725 | 1 | 1 | 1 |
| 4923-038 | 1726 | 1 | 1 | 1 |
| 4923-039 | 1727 | 1 | 1 | 1 |
| 4923-040 | 1728 | 1 | 1 | 1 |
| 4923-041 | 1769 | 1 | 1 | 1 |
| 4923-042 | 1770 | 1 | 1 | 1 |
| 4923-043 | 1771 | 1 | 1 | 1 |
| 4923-044 | 1772 | 1 | 1 | 1 |
| 4923-045 | 1773 | 1 | 1 | 1 |
| 4923-046 | 1774 | 1 | 1 | 1 |
| 4923-047 | 3025 | 1 | 1 | 1 |
| 4923-048 | 3028 | 1 | 1 | 1 |
| 4923-049 | 3026 | 1 | 1 | 1 |
| 4923-050 | 3027 | 1 | 1 | 1 |
| 4923-051 | 3197 | 1 | 1 | 1 |
| 4923-052 | 3198 | 1 | 1 | 1 |
| 4923-053 | 3199 | 1 | 1 | 1 |
| 4923-054 | 3200 | 1 | 1 | 1 |
| 4923-055 | 3205 | 1 | 1 | 0 |
| 4923-056 | 3206 | 1 | 1 | 1 |

| PATID | RANDOM<br>NUMBER | SAFETY | FAS | PP |
|----------|------------------|--------|-----|----|
| 4923-057 | 3207 | 1 | 1 | 1 |
| 4923-058 | 3208 | 1 | 1 | 1 |
| 4923-059 | 3273 | 1 | 1 | 1 |
| 4923-060 | 3274 | 1 | 1 | 1 |
| 4923-061 | 3275 | 1 | 1 | 1 |
| 4923-062 | 3276 | 1 | 1 | 1 |
| 4923-063 | 3277 | 1 | 1 | 1 |
| 4923-064 | 3278 | 1 | 1 | 1 |
| 4926-001 | 1521 | 1 | 1 | 1 |
| 4926-002 | 1522 | 1 | 1 | 1 |
| 4926-007 | 1527 | 1 | 1 | 1 |
| 4928-001 | 1273 | 1 | 1 | 1 |
| 4928-002 | 1274 | 1 | 1 | 1 |
| 4928-003 | 1275 | 1 | 1 | 1 |
| 4928-004 | 1276 | 1 | 1 | 1 |
| 4928-005 | 1277 | 1 | 1 | 1 |
| 4928-006 | 1278 | 1 | 1 | 1 |
| 4928-007 | 1279 | 1 | 1 | 1 |
| 4928-008 | 3033 | 1 | 1 | 1 |
| 4929-001 | 1433 | 1 | 1 | 1 |
| 4929-002 | 1434 | 1 | 1 | 1 |
| 4929-003 | 1435 | 1 | 1 | 1 |
| 4929-004 | 1436 | 1 | 1 | 1 |
| 4929-005 | 1437 | 1 | 1 | 1 |
| 4930-009 | 1665 | 1 | 1 | 0 |
| 4930-010 | 1666 | 1 | 1 | 1 |
| 4930-011 | 3040 | 1 | 1 | 1 |
| 4932-001 | 1265 | 1 | 1 | 1 |
| 4932-002 | 1266 | 1 | 1 | 1 |
| 4932-003 | 1267 | 1 | 1 | 1 |
| 4932-004 | 1268 | 1 | 1 | 1 |
| 4932-005 | 1269 | 1 | 1 | 1 |
| 4932-006 | 1270 | 1 | 1 | 1 |
| 4932-007 | 1271 | 1 | 1 | 1 |
| 4932-008 | 1272 | 1 | 1 | 1 |
| 4932-009 | 1681 | 1 | 1 | 1 |
| 4932-010 | 1682 | 1 | 1 | 1 |
| 4932-011 | 3041 | 1 | 1 | 1 |
| 4932-012 | 3042 | 1 | 1 | 1 |
| 4934-001 | 1609 | 1 | 1 | 1 |
| 4934-002 | 1610 | 1 | 1 | 1 |
| 4934-003 | 1612 | 1 | 1 | 1 |

| PATID | RANDOM<br>NUMBER | SAFETY | FAS | PP |
|----------|------------------|--------|-----|----|
| 4934-004 | 1611 | 1 | 1 | 1 |
| 4934-005 | 1613 | 1 | 1 | 1 |
| 4934-006 | 1614 | 1 | 1 | 1 |
| 4934-007 | 1615 | 1 | 1 | 1 |
| 4934-008 | 1616 | 1 | 1 | 1 |
| 4934-009 | 1713 | 1 | 1 | 1 |
| 4934-010 | 1714 | 1 | 1 | 1 |
| 4934-011 | 1715 | 1 | 1 | 1 |
| 4934-012 | 1716 | 1 | 1 | 1 |
| 4934-013 | 1717 | 1 | 1 | 1 |
| 4934-014 | 3045 | 1 | 1 | 1 |
| 4934-015 | 3046 | 1 | 0 | 0 |
| 4934-016 | 3047 | 1 | 1 | 1 |
| 4934-017 | 3048 | 1 | 1 | 1 |
| 4936-001 | 3081 | 1 | 1 | 1 |
| 4936-002 | 3082 | 1 | 1 | 1 |
| 4936-003 | 3083 | 1 | 1 | 1 |
| 4936-004 | 3084 | 1 | 1 | 1 |
| 4936-005 | 3157 | 1 | 1 | 1 |
| 4936-006 | 3158 | 1 | 1 | 1 |
| 4936-007 | 3159 | 1 | 1 | 1 |
| 4936-008 | 3160 | 1 | 1 | 1 |
| 4936-009 | 3225 | 1 | 1 | 1 |
| 4936-010 | 3226 | 1 | 1 | 1 |
| 4936-011 | 3227 | 1 | 1 | 1 |
| 4936-012 | 3228 | 1 | 1 | 1 |
| 4936-013 | 3229 | 1 | 1 | 1 |
| 4936-014 | 3230 | 1 | 1 | 1 |
| 4936-015 | 3231 | 1 | 1 | 1 |
| 4936-016 | 3232 | 1 | 1 | 1 |
| 4936-017 | 3281 | 1 | 1 | 1 |
| 4936-018 | 3282 | 1 | 1 | 1 |
| 4936-019 | 3283 | 1 | 1 | 1 |
| 4936-020 | 3284 | 1 | 1 | 1 |
| 4936-021 | 3285 | 1 | 1 | 1 |
| 4936-022 | 3286 | 1 | 1 | 1 |
| 4936-023 | 3287 | 1 | 1 | 1 |
| 4936-024 | 3288 | 1 | 1 | 1 |
| 4936-025 | 3313 | 1 | 1 | 1 |
| 4936-026 | 3314 | 1 | 1 | 1 |
| 4936-027 | 3315 | 1 | 1 | 1 |
| 4936-028 | 3316 | 1 | 1 | 1 |

| PATID | RANDOM<br>NUMBER | SAFETY | FAS | PP |
|----------|------------------|--------|-----|----|
| 4936-029 | 3325 | 1 | 1 | 1 |
| 4936-030 | 3326 | 1 | 1 | 1 |
| 4936-031 | 3327 | 1 | 1 | 1 |
| 4936-032 | 3328 | 1 | 1 | 1 |
| 4936-033 | 3333 | 1 | 1 | 1 |
| 4936-034 | 3334 | 1 | 1 | 1 |
| 4936-035 | 3335 | 1 | 1 | 1 |
| 4936-036 | 3336 | 1 | 1 | 1 |
| 4936-037 | 3337 | 1 | 1 | 1 |
| 4936-038 | 3338 | 1 | 1 | 1 |
| 4936-039 | 3339 | 1 | 1 | 1 |
| 4937-001 | 3137 | 1 | 1 | 1 |
| 4937-002 | 3138 | 1 | 1 | 1 |
| 4938-001 | 3141 | 1 | 1 | 1 |
| 4938-002 | 3142 | 1 | 1 | 0 |
| 4939-001 | 3217 | 1 | 1 | 1 |
| 4939-002 | 3218 | 1 | 1 | 1 |
| 4939-003 | 3219 | 1 | 1 | 1 |

Table 2: Dataset Assignment, Status: Hardlock Transfer, 'Issue' Patients (n = 184)

| PATID | RANDOM<br>NUMBER | SAFETY | FAS | PP |
|----------|------------------|--------|-----|----|
| 4905-001 | 1129 | 1 | 1 | 1 |
| 4905-002 | 1130 | 1 | 1 | 1 |
| 4905-003 | 1131 | 1 | 0 | 0 |
| 4905-004 | 1132 | 1 | 0 | 0 |
| 4905-005 | 1133 | 1 | 1 | 1 |
| 4905-006 | 1134 | 1 | 1 | 0 |
| 4905-007 | 1135 | 1 | 1 | 1 |
| 4905-008 | 1136 | 1 | 1 | 0 |
| 4905-011 | 1459 | 1 | 1 | 1 |
| 4905-012 | 1460 | 1 | 1 | 0 |
| 4909-003 | 1043 | 1 | 1 | 1 |
| 4909-004 | 1044 | 1 | 1 | 1 |
| 4909-005 | 1045 | 1 | 1 | 1 |
| 4909-006 | 1046 | 1 | 1 | 1 |
| 4909-007 | 1047 | 1 | 1 | 0 |
| 4909-008 | 1048 | 1 | 1 | 0 |
| 4909-009 | 1153 | 1 | 1 | 0 |
| 4909-010 | 1154 | 1 | 1 | 0 |
| 4909-013 | 1157 | 1 | 1 | 1 |
| 4909-014 | 1158 | 1 | 1 | 1 |
| 4909-020 | 1420 | 1 | 1 | 1 |
| 4909-021 | 1421 | 1 | 1 | 1 |
| 4909-022 | 1422 | 1 | 1 | 1 |
| 4909-023 | 1423 | 1 | 1 | 1 |
| 4909-024 | 1424 | 1 | 1 | 1 |
| 4909-025 | 1553 | 1 | 1 | 1 |
| 4909-026 | 1554 | 1 | 1 | 1 |
| 4909-027 | 1555 | 1 | 1 | 1 |
| 4909-028 | 1556 | 1 | 1 | 1 |
| 4909-029 | 1557 | 1 | 1 | 1 |
| 4909-030 | 1558 | 1 | 1 | 1 |
| 4909-031 | 1559 | 1 | 1 | 1 |
| 4909-032 | 1560 | 1 | 1 | 1 |
| 4909-033 | 1657 | 1 | 1 | 1 |
| 4909-034 | 1658 | 1 | 1 | 1 |
| 4909-035 | 1659 | 1 | 1 | 1 |
| 4910-001 | 1057 | 1 | 1 | 1 |
| 4910-002 | 1058 | 1 | 1 | 1 |
| 4910-003 | 1059 | 1 | 1 | 1 |
| 4910-004 | 1060 | 1 | 1 | 1 |

| PATID | RANDOM<br>NUMBER | SAFETY | FAS | PP |
|----------|------------------|--------|-----|----|
| 4910-005 | 1061 | 1 | 1 | 1 |
| 4910-006 | 1062 | 1 | 1 | 1 |
| 4910-007 | 1063 | 1 | 1 | 1 |
| 4910-008 | 1064 | 1 | 1 | 1 |
| 4910-009 | 1177 | 1 | 1 | 1 |
| 4910-010 | 1178 | 1 | 1 | 1 |
| 4910-011 | 1179 | 1 | 1 | 1 |
| 4910-012 | 1180 | 1 | 1 | 1 |
| 4910-013 | 1181 | 1 | 1 | 1 |
| 4910-014 | 1182 | 1 | 1 | 1 |
| 4910-015 | 1183 | 1 | 1 | 1 |
| 4910-016 | 1184 | 1 | 1 | 1 |
| 4910-017 | 1321 | 1 | 1 | 1 |
| 4910-018 | 1322 | 1 | 1 | 1 |
| 4910-019 | 1323 | 1 | 1 | 1 |
| 4910-020 | 1324 | 1 | 1 | 1 |
| 4910-021 | 1325 | 1 | 1 | 1 |
| 4910-022 | 1326 | 1 | 1 | 1 |
| 4910-023 | 1327 | 1 | 1 | 1 |
| 4910-024 | 1328 | 1 | 1 | 1 |
| 4910-025 | 1425 | 1 | 1 | 1 |
| 4910-026 | 1426 | 1 | 1 | 1 |
| 4910-027 | 1427 | 1 | 1 | 1 |
| 4910-028 | 1428 | 1 | 1 | 1 |
| 4910-029 | 1429 | 1 | 1 | 1 |
| 4910-030 | 1430 | 1 | 1 | 1 |
| 4910-031 | 1431 | 1 | 1 | 1 |
| 4910-032 | 1432 | 1 | 1 | 1 |
| 4910-033 | 1497 | 1 | 1 | 1 |
| 4910-034 | 1498 | 1 | 1 | 1 |
| 4910-035 | 1499 | 1 | 1 | 1 |
| 4910-036 | 1500 | 1 | 1 | 1 |
| 4910-037 | 1501 | 1 | 1 | 1 |
| 4910-038 | 1502 | 1 | 1 | 1 |
| 4910-039 | 1503 | 1 | 1 | 1 |
| 4910-040 | 1504 | 1 | 1 | 1 |
| 4910-041 | 1641 | 1 | 1 | 1 |
| 4910-042 | 1642 | 1 | 1 | 1 |
| 4910-043 | 1643 | 1 | 1 | 1 |
| 4910-044 | 1644 | 1 | 1 | 1 |
| 4910-045 | 1645 | 1 | 1 | 1 |
| 4911-001 | 1137 | 1 | 1 | 1 |

| PATID | RANDOM<br>NUMBER | SAFETY | FAS | PP |
|----------|------------------|--------|-----|----|
| 4911-002 | 1138 | 1 | 1 | 1 |
| 4911-003 | 1139 | 1 | 1 | 0 |
| 4911-004 | 1140 | 1 | 1 | 1 |
| 4911-005 | 1141 | 1 | 1 | 1 |
| 4917-001 | 1249 | 1 | 1 | 1 |
| 4917-002 | 1250 | 1 | 0 | 0 |
| 4917-003 | 1251 | 1 | 1 | 1 |
| 4918-001 | 1081 | 1 | 1 | 1 |
| 4918-002 | 1082 | 1 | 1 | 1 |
| 4918-003 | 1083 | 1 | 1 | 1 |
| 4918-004 | 1084 | 1 | 1 | 1 |
| 4918-005 | 1085 | 1 | 1 | 1 |
| 4918-006 | 1086 | 1 | 1 | 1 |
| 4918-007 | 1087 | 1 | 1 | 1 |
| 4918-008 | 1088 | 1 | 1 | 1 |
| 4918-009 | 1313 | 1 | 1 | 1 |
| 4918-010 | 1314 | 1 | 1 | 1 |
| 4918-011 | 1315 | 1 | 1 | 1 |
| 4918-012 | 1316 | 1 | 1 | 1 |
| 4918-013 | 1317 | 1 | 1 | 1 |
| 4918-014 | 1318 | 1 | 1 | 1 |
| 4918-018 | 1514 | 1 | 1 | 1 |
| 4921-001 | 1105 | 1 | 1 | 1 |
| 4921-003 | 1107 | 1 | 1 | 1 |
| 4921-004 | 1108 | 1 | 1 | 1 |
| 4921-005 | 1109 | 1 | 1 | 1 |
| 4921-006 | 1110 | 1 | 1 | 1 |
| 4921-007 | 1111 | 1 | 1 | 1 |
| 4921-008 | 1112 | 1 | 1 | 1 |
| 4921-009 | 1289 | 1 | 1 | 0 |
| 4921-010 | 1290 | 1 | 1 | 1 |
| 4921-014 | 1294 | 1 | 1 | 1 |
| 4921-015 | 1295 | 1 | 1 | 1 |
| 4921-017 | 1370 | 1 | 1 | 1 |
| 4921-018 | 1371 | 1 | 1 | 1 |
| 4921-019 | 1372 | 1 | 1 | 1 |
| 4921-026 | 1466 | 1 | 1 | 0 |
| 4921-028 | 1468 | 1 | 1 | 1 |
| 4921-030 | 1470 | 1 | 1 | 1 |
| 4921-031 | 1471 | 1 | 1 | 1 |
| 4921-032 | 1472 | 1 | 1 | 0 |
| 4921-033 | 1569 | 1 | 1 | 1 |

| PATID | RANDOM<br>NUMBER | SAFETY | FAS | PP |
|----------|------------------|--------|-----|----|
| 4921-034 | 1570 | 1 | 1 | 1 |
| 4921-035 | 1571 | 1 | 1 | 1 |
| 4921-036 | 1572 | 1 | 1 | 1 |
| 4921-037 | 1573 | 1 | 1 | 1 |
| 4921-038 | 1574 | 1 | 1 | 1 |
| 4921-040 | 1576 | 1 | 1 | 1 |
| 4921-041 | 1617 | 1 | 1 | 1 |
| 4921-042 | 1618 | 1 | 1 | 1 |
| 4921-043 | 1619 | 1 | 1 | 1 |
| 4921-044 | 1620 | 1 | 1 | 1 |
| 4921-045 | 1621 | 1 | 1 | 1 |
| 4921-046 | 1622 | 1 | 1 | 1 |
| 4921-047 | 1623 | 1 | 1 | 1 |
| 4921-051 | 1691 | 1 | 1 | 1 |
| 4921-052 | 1692 | 1 | 1 | 1 |
| 4921-053 | 1693 | 1 | 1 | 1 |
| 4921-054 | 1694 | 1 | 1 | 1 |
| 4923-001 | 1505 | 1 | 1 | 1 |
| 4923-002 | 1506 | 1 | 1 | 1 |
| 4923-003 | 1507 | 1 | 1 | 1 |
| 4923-004 | 1508 | 1 | 1 | 1 |
| 4923-005 | 1509 | 1 | 1 | 0 |
| 4923-006 | 1510 | 1 | 1 | 1 |
| 4923-007 | 1511 | 1 | 1 | 1 |
| 4923-008 | 1512 | 1 | 1 | 1 |
| 4923-009 | 1529 | 1 | 1 | 1 |
| 4923-010 | 1530 | 1 | 1 | 1 |
| 4923-011 | 1531 | 1 | 1 | 1 |
| 4923-012 | 1532 | 1 | 1 | 1 |
| 4923-013 | 1533 | 1 | 1 | 1 |
| 4923-014 | 1534 | 1 | 1 | 1 |
| 4923-015 | 1535 | 1 | 1 | 1 |
| 4923-016 | 1536 | 1 | 1 | 1 |
| 4923-017 | 1545 | 1 | 1 | 1 |
| 4923-018 | 1546 | 1 | 1 | 1 |
| 4923-019 | 1547 | 1 | 1 | 1 |
| 4923-020 | 1548 | 1 | 1 | 1 |
| 4923-021 | 1549 | 1 | 1 | 1 |
| 4923-022 | 1551 | 1 | 1 | 1 |
| 4923-023 | 1550 | 1 | 1 | 0 |
| 4923-024 | 1552 | 1 | 1 | 1 |
| 4923-025 | 1625 | 1 | 1 | 1 |

| PATID | RANDOM<br>NUMBER | SAFETY | FAS | PP |
|----------|------------------|--------|-----|----|
| 4923-026 | 1626 | 1 | 1 | 1 |
| 4923-027 | 1627 | 1 | 1 | 1 |
| 4923-028 | 1628 | 1 | 1 | 1 |
| 4923-029 | 1629 | 1 | 1 | 1 |
| 4926-003 | 1523 | 1 | 1 | 1 |
| 4926-004 | 1524 | 1 | 1 | 1 |
| 4926-005 | 1525 | 1 | 1 | 1 |
| 4926-006 | 1526 | 1 | 0 | 0 |
| 4930-001 | 1593 | 1 | 1 | 1 |
| 4930-002 | 1594 | 1 | 1 | 1 |
| 4930-003 | 1595 | 1 | 1 | 1 |
| 4930-004 | 1596 | 1 | 1 | 1 |
| 4930-005 | 1597 | 1 | 0 | 0 |
| 4930-006 | 1598 | 1 | 1 | 0 |
| 4930-007 | 1599 | 1 | 1 | 0 |
| 4930-008 | 1600 | 1 | 1 | 0 |
| 4931-001 | 1377 | 1 | 1 | 1 |
| 4931-002 | 1378 | 1 | 1 | 1 |

### 13.3 Table of Contents for Data Displays (Items of eCRF)

All items of the eCRF will be presented in individual participant data listings and in appropriate summary tables. Standard descriptive summary statistics will be calculated for continuous and semi-continuous variables (i.e., arithmetic mean, standard deviation, standard error of the mean, minimum value, lower quartile, median, upper quartile, maximum value, number of non-missing values). In addition, measures for skewness and kurtosis will be provided for suitable efficacy variables. Categorical data will be presented in frequency tables using counts and their associated percentages. Individual participant data listings will be presented per eCRF item and will be sorted appropriately. Summary tables will be displayed by treatment conditions and visit (if applicable). Where appropriate, the presentation will include changes from baseline. Semi-quantitative and quantitative efficacy data will be additionally visualized by boxplot diagrams. All standardized effect sizes (Mann-Whitney) will be visualized with their corresponding 95%-confidence intervals. All standard statistical tables will be generated applying the standard table layout of the validated statistical package TESTIMATE V6.5.14 (IDV Gauting). Associated meta-data and variable labels are finalized before unblinding All standard scientific figures are generated applying the standard figure layout of the validated scientific package SCIENCEGRAPH V4.9.39 (IDV Gauting).

KLIFO-013.05-A1.02

Data displays will be provided for the following analysis sets:

| Chapter Title | Analysis set |
|---|---|
| Study Patients | A: All patients randomized |
| Demographic and Other Baseline<br>Characteristics | B: Safety analysis set C: Full analysis set D: Per-protocol analysis set |
| Treatment Compliance | B: Safety analysis set C: Full analysis set D: Per-protocol analysis set |
| Visits | B: Safety analysis set C: Full analysis set D: Per-protocol analysis set |
| Analysis of Efficacy | C: Full analysis set D: Per-protocol analysis set |
| Analysis of Concomitant/ Supportive Therapies | B: Safety analysis set C: Full analysis set D: Per-protocol analysis set |
| Analysis of Safety | B: Safety analysis set |

# 13.3.1 Tables

# **Study Patients**

| Sections |
|---------------------------------|
| Disposition of Patients |
| End of Study / End of Treatment |
| Inclusion/Exclusion Criteria |
| Major Protocol Violations |
| Analysis Sets |

# **Demographic and Other Baseline Characteristics**

| Chapter Title |
|------------------------------------------------------------|
| Demography |
| Pregnancy Test |
| Medical History |
| Physical Examination / Vital Signs |
| Prior and Concomitant Medications |
| Time and Grading of Injury / Confirmatory Check of Grading |
| Supportive Therapy |
| VAS |
| FAAM |

# **Treatments**

| Chapter Title |
|---------------------------|
| Study Drug Administration |
| Compliance |

#### Visits

Chapter Title

Visits Intervals

# Efficacy Analysis

Chapter Title

VAS Pain on Passive Movement at Visits

AUC for VAS Pain on Passive Movement at Visits

VAS Pain at Rest at Visits

AUC for VAS Pain at Rest at Visits

Time to 50% Improvement for VAS Pain at Rest at Visits

Rescue Medication

# Concomitant/ Supportive Therapies

Chapter Title

Other Pain Medication

Supportive Therapy

**Concomitant Medications** 

# Safety Analysis

Chapter Title

Extent of Exposure

Adverse Events

Physical Examination / Vital Signs

# 13.3.2 Listings

# **Study Patients**

| Sections |
|---------------------------------|
| Disposition of Patients |
| End of Study / End of Treatment |
| Inclusion/Exclusion Criteria |
| Major Protocol Violations |
| Analysis Sets |

# **Demographic and Other Baseline Characteristics**

| Chapter Title |
|------------------------------------------------------------|
| Demography |
| Pregnancy Test |
| Medical History |
| Physical Examination / Vital Signs |
| Prior and Concomitant Medications |
| Time and Grading of Injury / Confirmatory Check of Grading |
| Supportive Therapy |
| VAS |
| FAAM |

## **Treatments**

| Chapter Title |
|---------------------------|
| Study Drug Administration |
| Compliance |

#### Visits

Chapter Title

Visits Intervals

## **Efficacy Analysis**

Chapter Title

VAS Pain on Passive Movement at Visits

AUC for VAS Pain on Passive Movement at Visits

VAS Pain at Rest at Visits

AUC for VAS Pain at Rest at Visits

Time to 50% Improvement for VAS Pain at Rest at Visits

Rescue Medication

## Concomitant/ Supportive Therapies

Chapter Title

Other Pain Medication

Supportive Therapy

Concomitant Medications

## Safety Analysis

Chapter Title

Extent of Exposure

Adverse Events

Physical Examination / Vital Signs

# 13.3.3 Figures

# Efficacy analysis

| Chapter Title | Type of Figure |
|---|---|
| VAS Pain on Passive Movement at Visits | Boxplots across all points in time (per group and visit); Means with standard deviation across all points in time (per group and visit); Standardized effect sizes (MW) with CI across all points in time (per group and visit) |
| AUC for VAS Pain on Passive Movement at Visits | Boxplots across all points in time (per group and follow-up visit); Means with standard deviation across all points in time (per group and follow-up visit); Standardized effect sizes (MW) with CI across all points in time (per group and follow-up visit); Scattergram for primary endpoint at Day 4 with regression lines (baseline VAS as covariate) |
| VAS Pain at Rest at Visits | Boxplots across all points in time (per group and visit); Means with standard deviation across all points in time (per group and visit); Standardized effect sizes (MW) with CI across all points in time (per group and visit) |
| AUC for VAS Pain at Rest at Visits | Boxplots across all points in time (per group and follow-up visit); Means with standard deviation across all points in time (per group and follow-up visit); Standardized effect sizes (MW) with CI across all points in time (per group and follow-up visit) |

| Time to 50% Improvement for VAS Pain at Rest at Visits | Kaplan Meier Curves per group. |
|---|---|
| Rescue Medication | Boxplots for Day 1 to 4 Totals per group, Boxplots for Day 1 to Final Day Totals per group; Standardized effect sizes (MW) for Day 1 to 4 Totals and Day 1 to Final Day Totals with CI per group. |

## 13.4 Clinical Trial Report (CTR) Specifications

## 13.4.1 Core CTR Specifications

The Core Clinical Trial Report (CTR) will be generated by means of the idv ICH-Study-Report-Manager V2.4.3 within the validated working environment at the department 'Clinical Research/ Biometry' in the institute IDV Data Analysis and Study Planning. The generation is based on the idv CTR template according to idv SOP KLIFO-16.04, the template being finalized before breaking the blind. The following specifications will apply to the CTR:

- Layout is DIN A4 format
- Body text font is Times New Roman 12 pt
- Language is American English (AE)
- CTR Structure is following the idv template according to idv SOP KLIFO-16.04
- CTR protocol sections are cited in original wording (unchanged or in past tense), the same applies to CTR SAP sections
- Scientific tables will be imported with full audit trail via validated pathway of module *idv-Tabellen/-Text*, remaining unchanged after import (original table)
- Scientific figures will be imported with full audit trail via validated pathway of module *idv Science-Graph-Tools*, remaining unchanged after import (original figure)
- Separate tables of content for core text, tables, and figures; generation by ICH-Study-Report-Manager V2.4.3
- CTR Versions:
  - Draft 0.1 (IDV Mock Report, generated before unblinding)
  - o Draft 1.0 (initial IDV CTR version after unblinding)
  - o Draft 1.X (follow-up CTR version after external review)
  - Draft to Final (IDV)
  - o Final (IDV)

# 13.4.2 Appendices:

- o Title pages generated according to title page of Core Report
- Appendix 1: Individual Patient Listing ('Non-Issue' Cases)
  - Listing of analysis data (validated XLI-export from TESTIMATE V6.5.14 analysis database with variable description by means of TESTIMATE V6.5.14 metadata)
- Appendix 2: Tables and Figures ('Non-Issue' Cases)
  - Tables will be imported with full audit trail via validated pathway of module idv-Tabellen/-Text, remaining unchanged after import (original scientific table)
  - Figures will be imported with full audit trail via validated pathway of module idv Science-Graph-Tools, remaining unchanged after import (original scientific figure)
- o Appendix 3: 'Issue" Cases
  - A. Individual Patient Listing (for specs see Appendix 1)
  - B. Tables and Figures (for specs see Appendix 2)
- Appendix 4: Listing of Original Raw Data Files (sas7bdat eCRF Domains) with variable description by means of latest version 4.0 of HE13226\_eCRF Specification (02 June 2020), sorting as shown in Table 3.

Table 3: Sorting of Individual Patient Data (sas 7bdat raw data)

| DOMAIN | DOMAIN TITLE | SORT BY |
|---|---|---|
| ADMIN | Study Drug<br>Administration | SEQNO |
| AE | Adverse Events | SEQID |
| AEGO | Adverse Events flags | |
| CCG | Confirmatory check of<br>Grading | VISITNO |
| COMMENTS<br>DA | Comments Rescue Medication Accountability | VISITNO |
| DIARYHO | Diary Handout | VISITNO |
| DM | Demography | S-SHIRS I |
| DOV | Visits | VISITNO |
| DS | Informed Consent | value emparer: RUSerTe(I) |
| EC | Exclusion Criteria | EXC |
| EOS | End of Study | |
| EOT | End of Treatment | |
| EVALP | Question to Patients | VISITNO |
| FAAM | Foot and Ankle Ability<br>Measure (FAAM) /<br>Activities of Daily Living | VISITNO |
| GDD | (ADL) Subscale Date of Confirmation of Grade 3 - Discontinuation of Treatment | |
| GRAD | Time and Grading of<br>Injury | VISITNO |
| IC | Inclusion Criteria | INC |
| LINK | Link list | |
| МН | Medical History | SEQNO |
| MHGO | Medical History flags | VISITNO |
| NA | Not Applicable | SEQNO |
| OPM | Other Pain Medications | STUDDCD |
| PARAC | Rescue Medication | STUDDCD |
| PCM | Prior and Concomitant<br>Medications | CMSEQ |

| DOMAIN | DOMAIN TITLE | SORT BY |
|---|---|---|
| PCMGO | Prior and Concomitant<br>Medications flags | |
| PE | Physical Examination | SEQNO |
| PEGO | Physical Examination flags | VISITNO |
| PREG<br>RAND | Pregnancy Test (only for<br>female patients with<br>childbearing potential)<br>Randomization | VISITNO |
| SUPT | Supportive Therapy | VISITNO |
| TAEC | Occurence of Adverse<br>Events | VISITNO |
| TCMC | Occurence of<br>Concomitant Medications | VISITNO |
| UNBLIND | Medical Code Broken | |
| VAS | Visual Analogue Scale | VISITNO |
| VS | Vital Signs | VISITNO |